# Replication of the POET-COPD Trial in Healthcare Claims Data

**DUPLICATE POET-COPD** 

August 10, 2021

#### 1. RCT Details

This section provides a high-level overview of an RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Tiotropium versus Salmeterol for the Prevention of Exacerbations of COPD (POET-COPD trial)

## 1.2 Intended aim(s)

The objective of the study is to assess the efficacy and safety of tiotropium, a long-acting anticholinergic (muscarinic antagonist) drug (LAMA) compared to salmeterol, a long-acting beta agonist (LABA) in patients with chronic obstructive pulmonary disease (COPD)

## 1.3 Primary endpoint for replication and RCT finding

Time to first COPD exacerbation

## 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

With a sample size of approximately 6800 patients (3400 in each arm), the trial will have 80% power to detect a 10% reduction in the risk of first exacerbation with tiotropium as compared with salmeterol, with a two-sided test for the null hypothesis of a hazard ratio of 1 at a significance level of 0.05

## 1.5 Trial estimate

HR = 0.83 (95% CI 0.77–0.90) comparing tiotropium to salmeterol (Vogelmeier et al., 2011, NEJM)

# 2. Person responsible for implementation of replication in Aetion

Helen Tesfaye, Pharm.D, ScM implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of design and analytic choices. All implementation steps are recorded, and implementation history is archived in the platform.

## 3. Data Source(s)

Optum Cliniformatics Data Mart, IBM MarketScan

# 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expediated review

# Design Diagram - POET-COPD TRIAL REPLICATION



## 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score matched retrospective cohort study design comparing tiotropium to salmeterol. The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of tiotropium or salmeterol inhalers (cohort entry date).

## 5.2 Important steps for cohort formation

New users (defined as no use in 180 days prior to index date) of an exposure and a comparator drug will be identified.

## 5.2.1 Eligible cohort entry date

Tiotropium inhaler was first approved by FDA for market availability on January 30, 2004, and salmeterol on September 15, 1998

- Optum: January 30, 2004 March 31, 2020 (end of data availability is December 31, 2020 but excluded data generated during COVID-19 pandemic)
- Marketscan: January 30, 2004 December 31, 2018 (end of data availability)

# 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

# 5.3 Flowchart of the study cohort assembly

| | OPT | UM | MARKE | TSCAN |
|---|---|---|---|---|
| | Less Excluded<br>Patients | Remaining<br>Patients | Less Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 79,335,559 | | 200,203,908 |
| Did not meet cohort entry criteria | -78,723,324 | 612,235 | -199,335,696 | 868,212 |
| Excluded due to insufficient enrollment | -87,210 | 525,025 | -98,266 | 769,946 |
| Excluded due to prior use of referent | -22,073 | 502,952 | -52,587 | 717,359 |
| Excluded due to prior use of exposure | -298,940 | 204,012 | -406,646 | 310,713 |
| Excluded because patient qualified in >1 exposure category | -164 | 203,848 | -292 | 310,421 |
| Excluded based on Missing/Unknown Age | 0 | 203,848 | 0 | 310,421 |
| Excluded based on Missing/Unknown Gender | -37 | 203,811 | 0 | 310,421 |
| Excluded based on Inclusion #1 - Age >=40 years old | -9,129 | 194,682 | -19,097 | 291,324 |
| Excluded based on Inclusion #2 - Diagnosis of COPD | -35,444 | 159,238 | -78,651 | 212,673 |
| Excluded based on Inclusion #4 - History of at least 1 COPD Exacerbation within the past year | -75,207 | 84,031 | -105,442 | 107,231 |
| Excluded based on Exclusion #2a - Asthma | -10,054 | 73,977 | -8,159 | 99,072 |
| Excluded based on Exclusion #2b - Severe cardiovascular or pulmonary disorders_V2 | -8,122 | 65,855 | -8,509 | 90,563 |
| Excluded based on Exclusion #3 - Patients with any respiratory infection or COPD exacerbation in the 4 weeks prior to visit 1 | -12,040 | 53,815 | -14,085 | 76,478 |
| Excluded based on Exclusion #5 - Salmeterol, Tiotropium containing inhaler use within 180 days* | -4,157 | 49,658 | -7,817 | 68,661 |
| Final cohort | | 49,658 | | 68,661 |

<sup>\*</sup> Additional exclusion criteria applied for replication

#### 6 Variables

## 6.1 Exposure-related variables:

### Study drug:

The study exposure of interest is initiation of tiotropium (LAMA). Initiation will be defined by no use of inhaled tiotropium during the prior 180 days before treatment initiation (washout period). Patients are required to be incident users with respect both exposure groups.

## **Comparator agents:**

Initiators of salmeterol inhaler defined as no use of inhaled salmeterol during the 180 days prior to index date

#### 6.2 Preliminary Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the default baseline covariate assessment period of 180 days prior to and including the index prescription date

Covariates listed above are a small subset of covariates that will ultimately be controlled in the design and analysis phase of the study. They are included in the preliminary assessment to determine the presence of adequate overlap between the two population of patients to proceed to the next phase of the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and initial power assessment and are listed in Table 1 (Appendix B).

# 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix A**):

- Primary outcome: Time to first COPD exacerbation
- Secondary outcome:
  - All-cause death

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted): Pneumonia

## 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analysis will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analysis, the follow-up will start the day after the initiation of tiotropium or salmeterol and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest,
- The date of end of continue registration in the database,
- End of the study period,
- Death,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (tiotropium or salmeterol) + a 60-day grace period,
- The date of switching from an exposure to comparator and vice versa,
- The date of switching to or initiation of other LAMA (excluding tiotropium) and other LABA (excluding salmeterol), LAMA/LABA, LABA/ICS, and LAMA/LABA/ICS combination inhalers.

For the ITT analyses, the censoring based on the switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

# 7 Initial Feasibility Analysis

Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1730/rwrs/71650">https://bwh-dope.aetion.com/projects/details/1730/rwrs/71650</a>
Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1732/rwrs/71648">https://bwh-dope.aetion.com/projects/details/1732/rwrs/71648</a>

<u>Date conducted:</u> 5/6/2021 (old version), 6/17/2021 (current) – In the current version, we removed the additional exclusion criteria "LABA, LAMA, or any combinations containing those (except study drugs) - 14 days washout period," which was applied in defining the cohort used in the old version.

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome.

- Complete study flowchart from Section 5.3
- Report patient characteristics by treatment group

| BEFORE MATCHING | | | | | | |
|---|---|---|---|---|---|---|
| | | Optum | | | Marketscan | |
| Variable | Referent -<br>Salmeterol | Exposure -<br>Tiotropium | Difference | Referent -<br>Salmeterol | Exposure -<br>Tiotropium | Difference |
| Number of patients | 1,077 | 48,581 | - (-, -) | 3,397 | 65,264 | - (-, -) |
| Age | | | | | | |
| mean (sd) | 69.31 (10.79) | 69.64 (9.85) | -0.34 (-0.99 <i>,</i><br>0.31) | 70.81 (10.79) | 68.26 (11.06) | 2.55 (2.18,<br>2.92) |
| median [IQR] | 70.00 [62.00,<br>77.50] | 70.00 [63.00,<br>77.00] | - (-, -) | 72.00 [63.00,<br>79.00] | 68.00 [60.00,<br>77.00] | - (-, -) |
| Gender | | | | | | |
| Male; n (%) | 511 (47.4%) | 21,601 (44.5%) | 3.0% (-0.1%,<br>6.0%) | 1,566 (46.1%) | 31,139 (47.7%) | -1.6% (-3.3%,<br>0.1%) |
| Female; n (%) | 566 (52.6%) | 26,980 (55.5%) | -3.0% (-6.0%,<br>0.1%) | 1,831 (53.9%) | 34,125 (52.3%) | 1.6% (-0.1%,<br>3.3%) |
| Combined comorbidity score, 180 days | | | | | | |
| mean (sd) | 2.37 (2.54) | 2.59 (2.56) | -0.22 (-0.37, -<br>0.06) | 1.75 (1.88) | 2.05 (2.14) | -0.31 (-0.37, -<br>0.24) |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 4.00] | - (-, -) | 1.00 [1.00, 3.00] | 1.00 [1.00, 3.00] | - (-, -) |

# Report summary parameters of study population

| FEASIBILITY FOR STUDY OUTCOME | | |
|---|---|---|
| | Optum | Marketscan |
| Variable | Value | Value |
| Number of patients in full cohort | 49,658 | 68,661 |
| Number of patients dropped as incomplete cases | 0 | 0 |
| Number of patients that did not begin follow-up | 57 | 72 |
| Number of patients in analytic cohort | 49,601 | 68,589 |
| Number of events | 11,400 | 15,086 |
| Number of person-years | 16,485.60 | 27,150.40 |
| Number of patients in group: Referent - Salmeterol | 1,073 | 3,389 |
| Number of patients in group: Exposure - Tiotropium | 48,528 | 65,200 |
| Risk per 1,000 patients | 229.83 | 219.95 |
| Rate per 1,000 person-years | 691.51 | 555.65 |

# Report median follow-up time by treatment group

| FOLLOW-UP TIME FOR STUDY OUTCOME Median Follow-Up Time (Days) [IQR] | | |
|---|---|---|
| Optum Marketscan | | |
| Patient Group | Median<br>Follow-Up Time<br>(Days) [IQR] | Median<br>Follow-Up<br>Time (Days)<br>[IQR] |
| Overall Patient Population | 88 [45, 140] | 88 [57, 148] |
| Referent - Salmeterol | 88 [56, 148] | 88 [73, 148] |
| Exposure - Tiotropium | 88 [45, 140] | 88 [56, 148] |

## Report reasons for censoring in the overall study population

| CENSORING REASONS FOR STUDY OUTCOME | | |
|---|---|---|
| | Optum | Marketscan |
| Overall | 49,601 | 68,589 |
| Death | 911 (1.8%) | 299 (0.4%) |
| Start of an additional exposure | 137 (0.3%) | 325 (0.5%) |
| End of index exposure | 19,798 (39.9%) | 29,908 (43.6%) |
| Specified date reached | 1,539 (3.1%) | 712 (1.0%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 3,174 (6.4%) | 7,894 (11.5%) |
| Switch to other LABA, LAMA + LABA/LAMA combo + LAMA/LABA/ICS combo + NH admissions Occurred | 12,687 (25.6%) | 14,442 (21.1%) |

#### 8 Initial Power Assessment

# Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1730/rwrs/71651">https://bwh-dope.aetion.com/projects/details/1730/rwrs/71651</a> Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1732/rwrs/71649">https://bwh-dope.aetion.com/projects/details/1732/rwrs/71649</a>

<u>Date conducted:</u> 5/4/2021 (old version), 6/17/2021 (current version) – In the current version, we removed the additional exclusion criteria "LABA, LAMA, or any combinations containing those (except study drugs) - 14 days washout period," which was applied in defining the cohort used in the old version.

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index.

| | Optum | Marketscan | Pooled |
|---------------------------------------|--------|------------|---------|
| Number of people matched | | | |
| Reference | 1073.0 | 3389.0 | 4462.0 |
| Exposure | 1073.0 | 3389.0 | 4462.0 |
| Risk per 1,000 patients | 229.8 | 220.0 | - |
| Rate per 1,000 person-years | 691.5 | 555.7 | |
| N of events | 11,400 | 15,086 | 26,486 |
| N of patients (both groups) at Step 1 | 49,658 | 68,661 | 118,319 |
| Risk per 1,000 patients | 229.57 | 219.72 | 223.85 |

| Superiority Analysis (Pooled) | |
|-------------------------------|-------------|
| Number of patients matched | |
| Reference | 4,462 |
| Exposed | 4,462 |
| Risk per 1,000 patients | 223.85 |
| Desired HR from RCT | 0.83 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 1997.6374 |
| Power | 0.986238897 |

| Superiority Analysis (Optum) | |
|------------------------------|-------------|
| Number of patients matched | |
| Reference | 1,073 |
| Exposed | 1,073 |
| Risk per 1,000 patients | 229.57 |
| Desired HR from RCT | 0.83 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 492.65722 |
| Power | 0.542994909 |

| Superiority Analysis (Marketscan) | |
|-----------------------------------|-------------|
| Number of patients matched | |
| Reference | 3,389 |
| Exposed | 3,389 |
| Risk per 1,000 patients | 219.72 |
| Desired HR from RCT | 0.83 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 1489.26216 |
| Power | 0.949012649 |

• Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: |
|-------------------------|--------------|----------------|
| Reviewed by FDA: | | Date reviewed: |
| Reasons for stopping | | |
| analysis (if required): | | |

## 9. Balance Assessment

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1730/rwrs/72136">https://bwh-dope.aetion.com/projects/details/1730/rwrs/72136</a>
Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1732/rwrs/72137">https://bwh-dope.aetion.com/projects/details/1732/rwrs/72137</a>

Date conducted: 7/6/2021

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

# • Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 0 (0%) | 0 (0%) | 0 (0%) |
| Death | 104 (1.19%) | 44 (1.01%) | 60 (1.38%) |
| Start of an additional exposure | 347 (3.98%) | 317 (7.27%) | 30 (0.69%) |
| End of Index Exposure | 5,180 (59.43%) | 2,735 (62.76%) | 2,445 (56.1%) |
| Specified date reached | 111 (1.27%) | 56 (1.28%) | 55 (1.26%) |
| End of patient enrollment | 1,133 (13%) | 485 (11.13%) | 648 (14.87%) |
| Switch to other LABA, LAMA + LABA/LAMA combo + LAMA/LABA/ICS combo + NH admissions Occurred | 1,841 (21.12%) | 721 (16.54%) | 1,120 (25.7%) |

# • Report follow-up time by treatment group.

| Patient Group | Optum<br>Median<br>Follow-Up Time<br>(Days) [IQR] | Marketscan<br>Median<br>Follow-Up Time<br>(Days) [IQR] |
|---|---|---|
| Overall Patient Population | 88 [83, 159] | 123 [88, 214] |
| Referent - Salmeterol | 88 [85, 154] | 125 [88, 195] |
| Exposure - Tiotropium | 88 [83, 169] | 122 [88, 226] |

# • Report overall risk of the primary outcome.

| | Optum | MarketScan | Pooled |
|-------------------------|--------|------------|--------|
| Risk per 1,000 patients | 229.57 | 219.72 | 223.85 |

## **10. Final Power Assessment**

Date conducted: 7/9/2021

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

| Superiority Analysis (Pooled) | |
|-------------------------------|-------------|
| Number of patients matched | |
| Reference | 4,358 |
| Exposed | 4,358 |
| Risk per 1,000 patients | 223.85 |
| Desired HR from RCT | 0.83 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 1951.0766 |
| Power | 0.984427581 |

| 1,073 |
|-------------|
| 1,073 |
| 229.57 |
| 0.83 |
| 0.05 |
| 492.65722 |
| 0.542994909 |
| an) |
| 3,285 |
| 3,285 |
| 219.72 |
| 0.83 |
| 0.05 |
| 1443.5604 |
| 0.942918994 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: |
|-------------------------|--------------|----------------|
| Reviewed by FDA: | | Date reviewed: |
| Reasons for stopping | | |
| analysis (if required): | | |

# Appendix A: COPD Exacerbation (primary outcome), All-cause mortality (secondary outcome)

#### **COPD Exacerbation**

Measured 1 day after drug initiation in primary diagnosis position specified below and inpatient care setting -

## **COPD** (Inpatient, Primary)

ICD-9 Diagnosis: 491.x, 492.x, 496 ICD-10 Diagnosis: J41.x, J42, J43.x, J44.x

#### OR

Measured 1 day after drug initiation in any diagnosis position specified below and inpatient and outpatient care setting AND steroid use within 14 days -

## **COPD** (Any care setting, Any position)

<u>ICD-9 Diagnosis</u>: 491.x, 492.x, 496 <u>ICD-10 Diagnosis</u>: J41.x, J42, J43.x, J44.x

AND

#### Corticosteroid systemic administration and/or oral prescription of --

- Prednisone
- Prednisolone
- Methylprednisolone
- Dexamethasone
- Hydrocortisone

\_\_\_\_\_

## **All-Cause Mortality**

Identified using the discharge status codes-

Optum-Inpatient/Outpatient

- 20 = EXPIRED
- 21 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 22 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 23 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 24 = EXPIRED TO BE DEFINED AT STATE LEVEL

- 25 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 26 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 27 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 28 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 29 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 40 = EXPIRED AT HOME (HOSPICE)
- 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE)
- 42 = EXPIRED PLACE UNKNOWN (HOSPICE)

#### Marketscan-Inpatient

- 20 Died
- 22 Died
- 23 Died
- 24 Died
- 25 Died
- 26 Died
- 27 Died
- 28 Died
- 29 Died
- 40 Other died status or Expired at home (Hospice claims only) (depends on year)
- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)
- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

# Appendix A

| | POIT-COPD trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|
| П | | | Please see the following Google drive for<br>further details or any missing information | |
| | | | https://drive.google.com/drive/folders/1W | Citatio |
| E | Trial details - intended 5 with label change - 2 we<br>DXPQSURE vs. COMPARISON | est run is | | Criteria Adequate mapping in claims |
| | Tiotropium 18 mcg once daily vs. Salmeterol hydrofluoroalkane 50 mcg twice daily | Tiotropium (Spiriva) vs. Salmeterol (Serevent) | | Intermediate mapping in claims |
| | Aim: To evaluate the effect of tiotropium compared to salmeterol on exacerbations of COPD | <u>Exposure</u> : Tiotropium <u>Reference</u> : Salmeterol | | |
| | PRIMARY QUITCOME | | | Poor mapping or cannot be<br>measured in claims |
| | | Measured 1 day after drug initiation in primary diagnosis position and inpatient care setting: | | |
| | | CDPD<br>ICD-9 Diagnosis: 491.x, 492.x, 496<br>ICD-10 Diagnosis: 141.x, 142, 143.x, 144.x | | |
| | | ICD-10 Diagnosis: I41.x, I42, I43.x, I44.x | | |
| | | OR | | |
| | | Measured 1 day after drug initiation in any diagnosis position and inpatient and outpatient | | |
| | | Measured 1 day after drug initiation in <u>any</u> diagnosis position and inpatient and outpatient<br>care setting AND steriod use within 14 days: | | |
| | Primary and point: Time to first COPD exacerbation within 1 year | cosp | | Can't be measured in claims but<br>not important for the analysis |
| | | ICD-9 Diagnosis: 491.x, 492.x, 496<br>ICD-10 Diagnosis: 141.x, 142, 143.x, 144.x | | not important for the analysis |
| | | AND | | |
| | | AND | | |
| | | Corticosteriod systemic administration and/or oral prescription of: | | |
| | | Carticonsterried volumes administration and/or oral prescription of - Predisione - Predisione - Ademyloge disclores - Decamination of - Predisione - Decamination oral | | |
| | | - Nethylprechiscione - Dexamethasone | | |
| | | - Hydrocortisone | 1 | |
| ь | Tiotropium 18 mcg once daily vs. Salmeterol hydroflouroali | iane 50 mcg twice daily | | |
| 1 | 40 years of age or older | Measured on the day of drug initiation Age >= 40 | i | |
| | | Measured from the start of all available data to the day of drug initiation in any diagnosis coultion and in the inpatient and outpatient care settine: | 1 | |
| | | | 1 | |
| 2 | Diagnosis of COPD | (109)<br>(CD-9 Disconnis: 491 v. 492 v. 495 | 1 | |
| | | CDPD<br>ICD-9 Diagnosis: 491.x, 492.x, 496<br>ICD-10 Diagnosis: 341.x, 342, 343.x, 344.x | i | |
| | | | 1 | |
| 3 | Post-bronchodilator FEV1 ≤ 70% of predicted normal and FEV1 ≤ 70% of FVC and a smoking history of ≥ 10 pack years | | 1 | |
| | | Measured 365 days prior to 28 days prior to drug initiation in primary diagnosis position<br>and inpatient care setting: | 1 | |
| | | | 1 | |
| | | COPD<br>ICD-9 Disensois: 491.x. 492.x. 496.0 | 1 | |
| | | ECD-9 Diagnosis: 491.x, 492.x, 496.0<br>ICD-10 Diagnosis: 141, 142.x, 143.x, 144.x | I | |
| | | or | i | |
| | | Measured 365 days prior to 28 days prior to drug initiation in any diagnosis maintain and | i | |
| | | Measured 365 days prior to 28 days prior to drug initiation in any diagnosis position and<br>inpatient and outpatient care setting AND steriod use within 14 days: | 1 | |
| 4 | History of at least 1 COPD exacerbation within the past year requiring treatment with antibiotics and/or systemic steriods and/o requiring hospitalization | ,<br>,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | i | |
| | | ICD-9 Diagnosis: 491.x, 492.x, 496.0<br>ICD-10 Diagnosis: 141.x, 142, 143.x, 144.x | 1 | |
| | | ICD-10 Diagnosis: 141.x, 142, 143.x, 144.x | i | |
| | | AND | | |
| | | Corticosteriod systemic administration and/or prescription - Predictions | 1 | |
| | | Corticonternod voltemic admirristration and/or prescription - Predisione - Predisione - Methylprednisclone | 1 | |
| ı | | - Metry prediscione | | |
| | | - Dexamethasone | | |
| | | - Dissamethasone<br>- Hydrocortisone | | |
| | DICLUSION CHITEINA | - Desamethasone<br>- Hydrocortisons | | |
| 1 | DICLUSION CHTDIAL Patients, with significant diseases other than COPD that would preclude puricipation in the trial or interpretation of the results are excluded. | - Dezamethiscore<br>- Hydrocortisone | | |
| 1 | DECUMENT WITH SIGNATURE AND STATE OF THE WORLD PRECISE SHEET STATE OF THE WORLD STATE OF | Decemenhations Hydrocontrions Indicators are carry prior to any monoting we say or only measurem any suggestion position and in the impatient and outpetient care setting: | | |
| 1 | ACCOMMENTAL AND ACCOMMENTAL AC | - Understanding - Pythoconstands - Pyth | | |
| 1 | DOUGHD CHEM Polish with applicant divisions other than COTO that would proclude participation in the trial of interpretation of the mode are schilder. | - Understanding - Pythoconstands - Pyth | | |
| 1 | According to the property diseases after that CFIS that would proclade participation in the half or interpretation of the made, or available. | Monamentum M | | |
| 1 | Occess with agellical disease, other than COTO that would procked participation in the total or expensation of the results<br>extended | - Understanding - Pythoconstands - Pyth | | |
| 1 | According to the second section of the control of t | And the continue of the contin | | |
| | Floriest with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | Indicational and a second seco | | |
| 1 | Foreign with graphest disease, other than COTO that would provided participation in the total or inseprendent of the resolu-<br>se annual of the control of the control of the control of the control of the resolu-<br>se annual or | And the contribution of th | | |
| | Floriest with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | Indicational and a second seco | | |
| | Floriest with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | months and the large-less and supplies are setting: Section 1.0 S | | |
| | Floriest with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | months and the large-less and supplies are setting: Section 1.0 S | | |
| | Floriest with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | months and the large-less and supplies are setting: Section 1.0 S | | |
| | Floriest with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | position and his largetist and application are setting: Section 1.00 per setting to the largetist and application are setting: Section 1.00 per setting to the largetist and section 1.00 per setting to the largetist and the lar | | |
| | Planets with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | months and the large-less and supplies are setting: Section 1.0 S | | |
| | Planets with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | Indicentification Application of the Section of Section (Section of Section | | |
| | Planets with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | Indicatoristics Indica | | |
| | Planets with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | Indicentification Application of the Section of Section (Section of Section | | |
| | Planets with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | Indicatoristics Indica | | |
| | Policies with a current diagnosis of withms, severe conditions clude disorders and set of systemic continuement medication as unabled. | John State Commission of the C | | |
| | Planets with a current dispress of arthms, were cardionaccide disorders and one of apparent continuement medication of the results. | Indicators can see a series prime and control of the series and see a series and seed and see a series and see a series and seed and see a series and seed and | | |
| 2 | Frames with a current diagnosis of arthms, seems cardiovascular disorders and use of systemic cardiocatemic modification at modification with a current diagnosis of arthms, seems cardiovascular disorders and use of systemic cardiocatemic modification at modification. | Indicators and STEP years as an extracting the stay is used, as the stay of th | | |
| | Frames with a current diagnosis of arthms, seems cardiovascular disorders and use of systemic cardiocatemic modification at modification with a current diagnosis of arthms, seems cardiovascular disorders and use of systemic cardiocatemic modification at modification. | Indicators and STEP years as an extracting the stay is used, as the stay of th | | |
| 2 | Frames with a current diagnosis of arthms, seems cardiovascular disorders and use of systemic cardiocatemic modification at modification with a current diagnosis of arthms, seems cardiovascular disorders and use of systemic cardiocatemic modification at modification. | months and the big-prime of any prime are setting: Manual To against and the big-prime and subprime are setting: Manual To against and the big-prime and subprime are setting: 100-100 primes 100 p | | |
| 2 | Follows with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders and one of systemic continuement medication at executive disorders. Protects with any respiratory infection or COSO essentiation* in the 4 weeks prior to the screening Visit (Visit 1) or during the con- in period. | indicates the second price of the second price | | |
| 2 | Frames with a current diagnosis of arthms, seems cardiovascular disorders and use of systemic cardiocatemic modification at modification with a current diagnosis of arthms, seems cardiovascular disorders and use of systemic cardiocatemic modification at modification. | indicates the second price of the second price | | |
| 2 | Follows with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders and one of systemic continuement medication at executive disorders. Protects with any respiratory infection or COSO essentiation* in the 4 weeks prior to the screening Visit (Visit 1) or during the con- in period. | months and the big-prime of any prime are setting: Manual To against and the big-prime and subprime are setting: Manual To against and the big-prime and subprime are setting: 100-100 primes 100 p | | |
| 2 | Follows with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders and one of systemic continuement medication at executive disorders. Protects with any respiratory infection or COSO essentiation* in the 4 weeks prior to the screening Visit (Visit 1) or during the con- in period. | indicates the second price of the second price | | |
| 2 | Follows with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders and one of systemic continuement medication at executive disorders. Protects with any respiratory infection or COSO essentiation* in the 4 weeks prior to the screening Visit (Visit 1) or during the con- in period. | Indicators of the State of the | | |
| 2 | Follows with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders and one of systemic continuement medication at executive disorders. Protects with any respiratory infection or COSO essentiation* in the 4 weeks prior to the screening Visit (Visit 1) or during the con- in period. | Indicatoristics Indica | | |
| 2 | Follows with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders and one of systemic continuement medication at executive disorders. Protects with any respiratory infection or COSO essentiation* in the 4 weeks prior to the screening Visit (Visit 1) or during the con- in period. | Indicators of the State of the | | |
| 2 | Follows with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders and one of systemic continuement medication at executive disorders. Protects with any respiratory infection or COSO essentiation* in the 4 weeks prior to the screening Visit (Visit 1) or during the con- in period. | Indicators and soft plan is not received, and so the students of the supplies of supplies of the supplies of supplies of the supplies of s | | |
| 2 | Follows with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders and one of systemic continuement medication at executive disorders. Protects with any respiratory infection or COSO essentiation* in the 4 weeks prior to the screening Visit (Visit 1) or during the con- in period. | indicatoristicism material of the September of Indicatoristicism of September of S | | |
| 2 | Foliates with a current diagnosis of arithms, severe condensecular disorders and one of systemic contributed and are severed and an extraction of the secular disorders and one of systemic contributed and are severed diagnosis of arithms, severe condensecular disorders and one of systemic contributed medication at entractive disorders and one of systemic contributed medication at each other systemic disorders and one of systemic contributed and one of sy | indicatoristicism material of the September of Indicatoristicism of September of S | | |
| 2 | Follows with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders with a current diagnosis of arithms, severe condensector disorders and one of systemic continuement medication at executive disorders and one of systemic continuement medication at executive disorders. Protects with any respiratory infection or COSO essentiation* in the 4 weeks prior to the screening Visit (Visit 1) or during the con- in period. | Indicatoristics Indica | | |
| 2 | Foliates with a current diagnosis of arithms, severe condensecular disorders and one of systemic contributed and are severed and an extraction of the secular disorders and one of systemic contributed and are severed diagnosis of arithms, severe condensecular disorders and one of systemic contributed medication at entractive disorders and one of systemic contributed medication at each other systemic disorders and one of systemic contributed and one of sy | indicatoristicism material of the September of Indicatoristicism of September of S | | |
| 2 | Foliates with a current diagnosis of arithms, severe condensecular disorders and one of systemic contributed and are severed and an extraction of the secular disorders and one of systemic contributed and are severed diagnosis of arithms, severe condensecular disorders and one of systemic contributed medication at entractive disorders and one of systemic contributed medication at each other systemic disorders and one of systemic contributed and one of sy | Indicators consists of the property of the constraint of the property of the constraint of the constra | | |
| 2 | Foliates with a current diagnosis of arithms, severe condensecular disorders and one of systemic contributed and are severed and an extraction of the secular disorders and one of systemic contributed and are severed diagnosis of arithms, severe condensecular disorders and one of systemic contributed medication at entractive disorders and one of systemic contributed medication at each other systemic disorders and one of systemic contributed and one of sy | indicatoristicism material of the September of Indicatoristicism of September of S | | |
| 3 | Foliates with a current diagnosis of arithms, severe condensecular disorders and one of systemic contributed and are severed and an extraction of the secular disorders and one of systemic contributed and are severed diagnosis of arithms, severe condensecular disorders and one of systemic contributed medication at entractive disorders and one of systemic contributed medication at each other systemic disorders and one of systemic contributed and one of sy | Indicators consists of the property of the constraint of the property of the constraint of the constra | | |



# Appendix B



# **UNMATCHED**

| | Referent - Salmeterol | OPTUM | | N | MARKETSCAN | | | POOLED | |
|---|---|---|---|---|---|---|---|---|---|
| Number of patients Calendar Time - Year of Initiation (2004 - 2020) | 1,077 | Exposure - Tiotropium<br>48,581 | | Referent - Salmeterol<br>3,397 | Exposure - Tiotropium<br>65,264 | | Referent - Salmeterol<br>4,474 | Exposure - Tiotropium<br>113,845 | |
| 2004-2006; n (%)<br>2007-2008; n (%) | 298 (27.7%)<br>104 (9.7%) | 2,777 (5.7%)<br>3,944 (8.1%) | 0.6173<br>0.0562 | 1,955 (57.6%)<br>404 (11.9%) | 9,783 (15.0%)<br>9,109 (14.0%) | 0.9881<br>-0.0626 | 2,253 (50.4%)<br>508 (11.4%) | 12,560 (11.0%)<br>13,053 (11.5%) | 0.945<br>-0.003 |
| 2009-2011; n (%)<br>2012-2015; n (%)<br>2012-2018: n (%) | 172 (16.0%)<br>157 (14.6%)<br>251 (23.3%) | 8,025 (16.5%)<br>13,877 (28.6%)<br>13,687 (28.2%) | -0.0136<br>-0.3452<br>-0.1122 | 545 (16.0%)<br>316 (9.3%)<br>177 (5.2%) | 17,106 (26.2%)<br>20,917 (32.0%)<br>8.349 (12.8%) | -0.2520<br>-0.5842<br>-0.2679 | 717 (16.0%)<br>473 (10.6%)<br>428 (9.6%) | 25,131 (22.1%)<br>34,794 (30.6%)<br>22,036 (19.4%) | -0.156<br>-0.510<br>-0.281 |
| 2016-2018; n (%)<br>2019-Mar. 2020; n (%) | 251 (23.3%)<br>95 (8.8%) | 6,271 (12.9%) | -0.1321 | 1// (5.2%) | 8,349 (12.8%) | -0.2679 | 95 (8.8%) | 6,271 (12.9%) | -0.132 |
| DMG - Age<br>mean (sd) | 69.31 (10.79) | 69.64 (9.85) | -0.0319 | 70.81 (10.79) | 68.26 (11.06) | 0.2334 | 70.45 (10.79) | 68.85 (10.56) | 0.150 |
| median [ICR] DMG - Gender | 70.00 [62.00, 77.50]<br>511 (47.4%) | 70.00 [63.00, 77.00] | 0.0000 | 72.00 [63.00, 79.00] | 68.00 [60.00, 77.00] | -0.0321 | 71.52 (10.79) | 68.85 (10.56)<br>52.740 (46.3%) | 0.250 |
| Male; n (%)Female; n (%) DMG - Geographic region | 511 (47.4%)<br>566 (52.6%) | 21,601 (44.5%)<br>26,980 (55.5%) | -0.0582 | 1,566 (46.1%)<br>1,831 (53.9%) | 31,139 (47.7%)<br>34,125 (52.3%) | 0.0321 | 2,077 (46.4%) 2,397 (53.6%) | 61,105 (53.7%) | -0.002 |
| Northeast; n (%)South; n (%) | 100 (9.3%)<br>385 (35.7%) | 5,118 (10.5%)<br>22,458 (46.2%) | -0.0402<br>-0.2148 | 351 (10.3%)<br>845 (24.9%) | 10,691 (16.4%)<br>23,650 (36.2%) | -0.1801<br>-0.2472 | 451 (10.1%)<br>1,230 (27.5%) | 15,809 (13.9%)<br>46,108 (40.5%) | -0.117<br>-0.277 |
| North Central; n (%)<br>West; n (%) | 278 (25.8%)<br>314 (29.2%) | 10,162 (20.9%)<br>10,843 (22.3%) | 0.1160<br>0.1583 | 1,108 (32.6%)<br>1,093 (32.2%) | 23,003 (35.2%)<br>7,920 (12.1%) | -0.0549<br>0.4989 | 1,386 (31.0%)<br>1,407 (31.4%) | 33,165 (29.1%)<br>18,763 (16.5%) | 0.041<br>0.355 |
| DRS - Combined comorbidity score, 180 daysmean [sd] | 2.37 (2.54) | 2.59 (2.56) | -0.0863<br>0.0000 | 1.75 (1.88) | 2.05 (2.14) | -0.1489<br>0.0000 | 1.90 (2.06)<br>1.24 (2.06) | 2.28 (2.33)<br>1.43 (2.33) | -0.173<br>-0.086 |
| median [IQR] DRS - Frailty Score: Empirical Version (mean)mean [xd] | 2.00 [1.00, 3.00]<br>0.21 (0.07) | 2.00 [1.00, 4.00]<br>0.22 (0.07) | -0.1429 | 1.00 [1.00, 3.00]<br>0.19 (0.06) | 0.20 (0.07) | -0.1534 | 0.19 (0.06) | 0.21 (0.07) | -0.307 |
| median [IQR] | 0.19 [0.16, 0.24] | 0.20 [0.16, 0.25] | -0.1429 | 0.18 [0.14, 0.22] | 0.19 [0.15, 0.23] | -0.1534 | 0.18 (0.06) | 0.19 (0.07) | -0.153 |
| PLM - Smoking; n (%) PLM - Pneumonia; n (%) | 304 (28.2%)<br>121 (11.2%) | 20,039 (41.2%)<br>6,244 (12.9%) | -0.2757<br>-0.0522<br>0.0397 | 328 (9.7%)<br>361 (10.6%) | 14,153 (21.7%)<br>8,855 (13.6%) | -0.3344 | 632 (14.1%)<br>482 (10.8%)<br>232 (5.2%) | 34,192 (30.0%)<br>15,099 (13.3%) | -0.391 |
| PLM - Alpha-1 antitrypsin def/Pneumoconioses & other lung disease/Pul fibrosis; n (%) PLM - Oxygen usage; n (%) PLM - Respiratory arrest/dependence on oxygen ; n (%) | 79 (7.3%)<br>155 (14.4%)<br>129 (12.0%) | 3,040 (6.3%)<br>7,652 (15.8%)<br>7,778 (16.0%) | -0.0391<br>-0.1155 | 153 (4.5%)<br>588 (17.3%)<br>227 (6.7%) | 3,648 (5.6%)<br>10,345 (15.9%)<br>7,027 (10.8%) | -0.0503<br>0.0376<br>-0.1455 | 743 (16.6%)<br>356 (8.0%) | 6,688 (5.9%)<br>17,997 (15.8%)<br>14.805 (13.0%) | -0.031<br>0.022<br>-0.164 |
| PLM - CIPAP/BIPAP use; n (%) PLM - Pulmonary rehabilitation ; n (%)* | 63 (5.8%)<br>7 (0.6%) | 3,294 (6.8%)<br>341 (0.7%) | -0.0412<br>-0.0124 | 132 (3.9%)<br>9 (0.3%) | 5,015 (7.7%)<br>470 (0.7%) | -0.1631<br>-0.0567 | 195 (4.4%)<br>016 (0.4%) | 8,309 (7.3%)<br>811 (0.7%) | -0.124<br>-0.041 |
| PLM - Moderate COPD exacerbation - [Count with 365 to 181 days before CED]*mean [sd] | 1.67 (4.35) | 2.72 (6.59) | -0.1881<br>-0.0752 | 1.53 (3.65) | 1.65 (3.78) | -0.0323<br>-0.0188 | 1.56 (3.83)<br>0.06 (3.83) | 2.11 (5.17)<br>0.27 (5.17) | -0.121<br>-0.046 |
| median [IQR] PLM - Moderate COPD exacerbation - [Count 180 to 31 days before CED]*mean [ud] | 0.00 [0.00, 1.14]<br>1.72 (3.96) | 0.42 [0.00, 2.57] | -0.1312 | 0.08 [0.00, 1.23]<br>1.29 (2.41) | 0.15 [0.00, 1.62] | -0.0188 | 1.39 (2.86) | 1.77 (3.44) | -0.120 |
| median [ICR] PLM - Moderate COPD exacerbation - [Count with 30 days to CED]* | 0.64 [0.01, 1.82] | 0.88 [0.13, 2.45] | -0.0573 | 0.53 [0.00, 1.35] | 0.61 [0.00, 1.66] | -0.0327 | 0.56 (2.86) | 0.73 (3.44) | -0.054 |
| mean (sd)median (ICR) | 0.29 (1.12)<br>0.00 [0.00, 0.00] | 0.30 (1.11)<br>0.00 [0.00, 0.00] | -0.0090<br>0.0000 | 0.16 (0.53)<br>0.00 [0.00, 0.00] | 0.21 (0.65)<br>0.00 [0.00, 0.00] | -0.0843<br>0.0000 | 0.19 (0.72)<br>0.00 (0.72) | 0.25 (0.88)<br>0.00 (0.88) | -0.075<br>0.000 |
| PLM - Moderate exacerbations >= 1 in 365 days before CED; n (%) PLM - Moderate exacerbations >= 2 in 365 days before CED; n (%) PLM - Swere CPD; near certainion, (County this 365 to 184) days before CED!* | 864 (80.2%)<br>576 (53.5%) | 40,971 (84.3%)<br>31,738 (65.3%) | -0.1075<br>-0.2420 | 2,520 (74.2%)<br>1,612 (47.5%) | 51,102 (78.3%)<br>35,919 (55.0%) | -0.0965<br>-0.1505 | 3,384 (75.6%)<br>2,188 (48.9%) | 92,073 (80.9%)<br>67,657 (59.4%) | -0.129<br>-0.212 |
| mean (sd) | 0.04 (0.20) | 0.07 (0.29)<br>0.00 [0.00, 0.00] | -0.1204<br>0.0000 | 0.06 (0.25)<br>0.00 [0.00, 0.00] | 0.07 (0.26) | -0.0392<br>0.0000 | 0.06 (0.24)<br>0.00 (0.24) | 0.07 (0.27)<br>0.00 (0.27) | -0.039<br>0.000 |
| PLM - Severe COPD exacerbation - [Count with 180 to 31 days before CED] *mean (sd) | 0.06 (0.26) | 0.06 (0.24) | 0.0000 | 0.06 (0.22) | 0.06 (0.21) | 0.0000 | 0.06 (0.23) | 0.06 (0.22) | 0.000 |
| median [IQR] PLM - Severe COPD exacerbation - [Count with 30 days lookback] *mean [kd] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.23) | 0.00 (0.22) | 0.000 |
| mean (sd)median (ICR) PLM - Severe exacerbations >=1 in 365 days before CED; n (%) | 0.01 (0.09)<br>0.00 [0.00, 0.00]<br>106 (9.8%) | 0.01 (0.10)<br>0.00 [0.00, 0.00]<br>6,395 (13.2%) | 0.0000 | 0.01 (0.06)<br>0.00 [0.00, 0.00]<br>428 (12.6%) | 0.01 (0.08)<br>0.00 [0.00, 0.00]<br>9,050 (13.9%) | 0.0000 | 0.01 (0.07)<br>0.00 (0.07)<br>534 (11.9%) | 0.01 (0.09)<br>0.00 (0.09)<br>15,445 (13.6%) | 0.000 |
| PLM - Severe exacerbations >= 2 in 365 days before CED ; n (%) PLM - GOLD C/D Status ; n (%) | 15 (1.4%)<br>437 (40.6%) | 1,226 (2.5%)<br>26,005 (53.5%) | -0.0796<br>-0.2606 | 66 (1.9%)<br>1,613 (47.5%) | 1,138 (1.7%)<br>35,581 (54.5%) | 0.0150<br>-0.1404 | 081 (1.8%)<br>2,050 (45.8%) | 2,364 (2.1%)<br>61,586 (54.1%) | -0.022<br>-0.167 |
| PRX - LABA (except salmeterol) inhalers; n (%) | 62 (5.8%)<br>14 (1.3%) | 847 (1.7%)<br>440 (0.9%) | 0.2171 | 195 (5.7%)<br>14 (0.4%) | 2,276 (3.5%) 520 (0.8%) | 0.1052 | 257 (5.7%)<br>028 (0.6%) | 3,123 (2.7%)<br>960 (0.8%) | 0.150 |
| PRX - LAMA (except tiotropium) inhalers; n (%) * PRX - ICS only inhalers; n (%) * PRX - LABA/LAMA inhaler use: n (%) * | 14 (1.5%)<br>416 (38.6%)<br>17 (1.6%) | 8,938 (18.4%)<br>503 (1.0%) | 0.4591 | 14 (U.4%)<br>1,638 (48.2%)<br>2 (0.1%) | 14,424 (22.1%)<br>206 (0.3%) | 0.5683 | 2,054 (45.9%)<br>019 (0.4%) | 23,362 (20.5%)<br>709 (0.6%) | 0.560 |
| PRX - LABA/ICS inhaler use; n (%) PRX - COPD Maintenance therapy inhalers; n (%) | 45 (4.2%)<br>126 (11.7%) | 11,055 (22.8%)<br>12,434 (25.6%) | -0.5657<br>-0.3627 | 107 (3.1%)<br>236 (6.9%) | 14,588 (22.4%)<br>13,496 (20.7%) | -0.6045<br>-0.4084 | 152 (3.4%)<br>362 (8.1%) | 25,643 (22.5%)<br>25,930 (22.8%) | -0.593<br>-0.415 |
| PRX - SAMA inhaler use; n (%) PRX - SABA use; n (%) | 108 (10.0%)<br>523 (48.6%) | 2,469 (5.1%)<br>25,017 (51.5%) | 0.1863<br>-0.0580 | 624 (18.4%)<br>1,562 (46.0%) | 3,835 (5.9%)<br>31,659 (48.5%) | 0.3898<br>-0.0501 | 732 (16.4%)<br>2,085 (46.6%) | 6,304 (5.5%)<br>56,676 (49.8%) | 0.355<br>-0.064 |
| PRX - SABA/SAMA use; n (%) PRX - Antibiotics treatment (180 days to 31 days before CED); n (%) | 243 (22.6%)<br>512 (47.5%) | 7,839 (16.1%)<br>24,200 (49.8%) | 0.1651<br>-0.0460<br>0.0562 | 839 (24.7%)<br>1,697 (50.0%) | 10,570 (16.2%)<br>34,160 (52.3%) | 0.2119<br>-0.0460<br>-0.0288 | 1,082 (24.2%)<br>2,209 (49.4%) | 18,409 (16.2%)<br>58,360 (51.3%) | -0.038 |
| PRX - Antibiotics treatment (30 days to CED); n (%) PRX - Systemic Corticosteroids (with CPT) use (180 to 31 days before CED); n (%) PRX - Systemic Corticosteroids (with CPT) use (30 days to CED); n (%) | 152 (14.1%)<br>539 (50.0%)<br>102 (9.5%) | 5,931 (12.2%)<br>25,127 (51.7%)<br>3.369 (6.9%) | -0.0340<br>0.0949 | 458 (13.5%)<br>1,638 (48.2%)<br>384 (11.3%) | 9,458 (14.5%)<br>32,585 (49.9%)<br>5,550 (8.5%) | -0.0288<br>-0.0340<br>0.0939 | 610 (13.6%)<br>2,177 (48.7%)<br>486 (10.9%) | 15,389 (13.5%)<br>57,712 (50.7%)<br>8,919 (7.8%) | 0.003<br>-0.040<br>0.107 |
| PRX - Roflumillast; n (%) * | 7 (0.6%) | 378 (0.8%) | -0.0240 | 5 (0.1%) | 487 (0.7%) | -0.0952 | 012 (0.3%) | 865 (0.8%) | -0.068 |
| CVD - Unstable angina /Mi ; n (%) CVD - Stable Angina ; n (%) | 86 (8.0%)<br>46 (4.3%) | 4,729 (9.7%)<br>2,338 (4.8%) | -0.0599<br>-0.0240 | 223 (6.6%)<br>95 (2.8%) | 4,791 (7.3%)<br>2,405 (3.7%) | -0.0275<br>-0.0508 | 309 (6.9%)<br>141 (3.2%) | 9,520 (8.4%)<br>4,743 (4.2%) | -0.056<br>-0.053 |
| CVD - Any Heart failure (HF); n (%) CVD - Atrial fibrillation; n (%) CVD - Other dysrythmias ; n (%)* | 183 (17.0%)<br>144 (13.4%)<br>191 (17.7%) | 9,631 (19.8%)<br>6,877 (14.2%)<br>8,444 (17.4%) | -0.0723<br>-0.0232<br>0.0079 | 518 (15.2%)<br>393 (11.6%)<br>352 (10.4%) | 11,652 (17.9%)<br>8,538 (13.1%)<br>9,481 (14.5%) | -0.0727<br>-0.0456<br>-0.1244 | 701 (15.7%)<br>537 (12.0%)<br>543 (12.1%) | 21,283 (18.7%)<br>15,415 (13.5%)<br>17,925 (15.7%) | -0.080<br>-0.045<br>-0.104 |
| CVD - Valve disorder: n (%) CVD - Implantable cardioverter defibrillator ; n (%)* | 34 (3.2%)<br>14 (1.3%) | 1,741 (3.6%)<br>951 (2.0%) | -0.0221<br>-0.0550 | 74 (2.2%)<br>32 (0.9%) | 1,841 (2.8%)<br>961 (1.5%) | -0.0384<br>-0.0551 | 108 (2.4%)<br>046 (1.0%) | 3,582 (3.1%)<br>1,912 (1.7%) | -0.043<br>-0.061 |
| CVD - CABG/PCI; n (%) CVD - Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 74 (6.9%)<br>270 (25.1%) | 4,336 (8.9%)<br>13,906 (28.6%) | -0.0742<br>-0.0790 | 139 (4.1%)<br>704 (20.7%) | 3,428 (5.3%)<br>17,219 (26.4%) | -0.0567<br>-0.1346 | 213 (4.8%)<br>974 (21.8%) | 7,764 (6.8%)<br>31,125 (27.3%) | -0.086<br>-0.128 |
| CVD - Stroke/f1A ; n (%) CVD - Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) | 60 (5.6%)<br>112 (10.4%) | 2,727 (5.6%)<br>6,337 (13.0%)<br>26,282 (54.1%) | 0.0000<br>-0.0810<br>-0.1243 | 169 (5.0%)<br>218 (6.4%)<br>703 (20.7%) | 3,400 (5.2%)<br>5,918 (9.1%)<br>22,385 (34.3%) | -0.0091<br>-0.1011<br>-0.3082 | 229 (5.1%)<br>330 (7.4%)<br>1.219 (27.2%) | 6,127 (5.4%)<br>12,255 (10.8%)<br>48,667 (42.7%) | -0.013<br>-0.118 |
| CVD - Hyperlipidemia ; n (%) CVD - Hypertension; n (%) | 516 (47.9%)<br>695 (64.5%) | 33,432 (68.8%) | -0.1243 | 1,384 (40.7%) | 22,385 (34.3%)<br>33,730 (51.7%) | -0.3082 | 2,079 (46.5%) | 48,667 (42.7%)<br>67,162 (59.0%) | -0.329<br>-0.252 |
| CRX - ACEI or ARB; n (%) CRX - Mineralocorticoid receptor antagonist ; n (%) | 457 (42.4%)<br>44 (4.1%) | 22,139 (45.6%)<br>2,041 (4.2%) | -0.0645<br>-0.0050 | 1,444 (42.5%)<br>161 (4.7%) | 29,179 (44.7%)<br>3,176 (4.9%) | -0.0444<br>-0.0094 | 1,901 (42.5%)<br>205 (4.6%) | 51,318 (45.1%)<br>5,217 (4.6%) | -0.052<br>0.000 |
| CRX - Loop or Thiazide diuretics; n (%) CRX - Statins and other lipid lowering agents; n (%) | 374 (34.7%)<br>487 (45.2%) | 16,506 (34.0%)<br>25,485 (52.5%)<br>17,833 (36.7%) | 0.0147<br>-0.1464 | 1,379 (40.6%)<br>1,511 (44.5%) | 23,473 (36.0%)<br>32,717 (50.1%)<br>23,987 (36.8%) | 0.0947<br>-0.1123 | 1,753 (39.2%)<br>1,998 (44.7%)<br>1,299 (29.0%) | 39,979 (35.1%)<br>58,202 (51.1%) | 0.085<br>-0.128 |
| CRX - Beta blockers; n (%) CRX - CCB and other antihypertensives; n (%) CRX - Digoxin; n (%)* | 342 (31.8%)<br>336 (31.2%)<br>52 (4.8%) | 17,833 (36.7%)<br>14,658 (30.2%)<br>1,689 (3.5%) | -0.1034<br>0.0217<br>0.0652 | 957 (28.2%)<br>1,148 (33.8%)<br>307 (9.0%) | 23,987 (36.8%)<br>19,244 (29.5%)<br>3,742 (5.7%) | -0.1844<br>0.0926<br>0.1267 | 1,299 (29.0%)<br>1,484 (33.2%)<br>359 (8.0%) | 41,820 (36.7%)<br>33,902 (29.8%)<br>5,431 (4.8%) | -0.164<br>0.073<br>0.131 |
| CRX - Nitrates; n (%)* | 100 (9.3%) | 4,486 (9.2%) | 0.0035 | 431 (12.7%) | 7,249 (11.1%) | 0.0494 | 531 (11.9%) | 11,735 (10.3%) | 0.051 |
| OCM - Type 1 or 2 DM; n (%) OCM - Occurrence of Diabetic retinopathy/nephropathy/neuropathy; n (%)* | 290 (26.9%)<br>91 (8.4%) | 13,869 (28.5%)<br>5,084 (10.5%) | -0.0358<br>-0.0718 | 681 (20.0%)<br>127 (3.7%) | 15,497 (23.7%)<br>3,524 (5.4%) | -0.0896<br>-0.0816 | 971 (21.7%)<br>218 (4.9%) | 29,366 (25.8%)<br>8,608 (7.6%) | -0.096<br>-0.112 |
| OCM - Hypertensive nephropathy; n (%)* OCM - Hypotension; n (%)* | 82 (7.6%)<br>42 (3.9%) | 4,127 (8.5%)<br>2,601 (5.4%) | -0.0331<br>-0.0713<br>-0.0180 | 100 (2.9%)<br>77 (2.3%) | 2,758 (4.2%)<br>2,518 (3.9%) | -0.0703<br>-0.0924<br>0.0000 | 182 (4.1%)<br>119 (2.7%)<br>088 (2.0%) | 6,885 (6.0%)<br>5,119 (4.5%)<br>2,576 (2.3%) | -0.087<br>-0.097<br>-0.021 |
| OCM - Hyperkalemia; n (%)* OCM - CKD II, III, or IV; n (%) OCM - HO/PD/SRD; n (%)* | 29 (2.7%)<br>94 (8.7%)<br>16 (1.5%) | 1,448 (3.0%)<br>5,205 (10.7%)<br>510 (1.0%) | -0.0180<br>-0.0676<br>0.0450 | 59 (1.7%)<br>80 (2.4%)<br>35 (1.0%) | 1,128 (1.7%)<br>3,244 (5.0%)<br>849 (1.3%) | -0.1381<br>-0.0281 | 088 (2.0%)<br>174 (3.9%)<br>051 (1.1%) | 2,576 (2.3%)<br>8,449 (7.4%)<br>1,359 (1.2%) | -0.021<br>-0.152<br>-0.009 |
| OCM - Osteoporosis; n (%) OCM - Steep agnes; n (%) | 135 (12.5%)<br>139 (12.9%) | 6,026 (12.4%)<br>7,636 (15.7%) | 0.0030 | 473 (13.9%)<br>236 (6.9%) | 6,609 (10.1%)<br>8,922 (13.7%) | 0.1171 | 608 (13.6%)<br>375 (8.4%) | 12,635 (11.1%)<br>16,558 (14.5%) | 0.076 |
| OCM - Fractures ; n (%) OCM - Other Arthritis, Arthropathies and Musculoskeletal Pain ; n (%) | 68 (6.3%)<br>463 (43.0%) | 3,465 (7.1%)<br>22,638 (46.6%) | -0.0320<br>-0.0724 | 218 (6.4%)<br>1,073 (31.6%) | 4,379 (6.7%)<br>25,228 (38.7%) | -0.0121<br>-0.1491 | 286 (6.4%)<br>1,536 (34.3%) | 7,844 (6.9%)<br>47,866 (42.0%) | -0.020<br>-0.159 |
| OCM - Dorsopathies; n (%) OCM - Gout (acute/chronic); n (%)* | 308 (28.6%)<br>7 (0.6%) | 16,451 (33.9%)<br>562 (1.2%) | -0.1145<br>-0.0636<br>-0.0778 | 671 (19.8%)<br>45 (1.3%) | 16,991 (26.0%)<br>799 (1.2%) | -0.1480<br>0.0090<br>-0.0135 | 979 (21.9%)<br>052 (1.2%)<br>021 (0.5%) | 33,442 (29.4%)<br>1,361 (1.2%)<br>837 (0.7%) | -0.172<br>0.000<br>-0.026 |
| OCM - Hyperthyroldism; n (%)* OCM - Hypothyroldism; n (%)* OCM - VTE; n (%)* | 3 (0.3%)<br>99 (9.2%)<br>40 (3.7%) | 420 (0.9%)<br>4,864 (10.0%)<br>1,870 (3.8%) | -0.0272<br>-0.0053 | 18 (0.5%)<br>217 (6.4%)<br>113 (3.3%) | 417 (0.6%)<br>5,362 (8.2%)<br>2,558 (3.9%) | -0.0692<br>-0.0322 | 316 (7.1%)<br>153 (3.4%) | 10,226 (9.0%) | -0.070<br>-0.027 |
| OCM - GERD ; n (%) OCM - Cancer ; n (%) | 203 (18.8%)<br>150 (13.9%) | 10,528 (21.7%)<br>6,452 (13.3%) | -0.0722<br>0.0175 | 244 (7.2%)<br>369 (10.9%) | 6,858 (10.5%)<br>7,334 (11.2%) | -0.1164<br>-0.0096 | 447 (10.0%)<br>519 (11.6%) | 17,386 (15.3%)<br>13,786 (12.1%) | -0.160<br>-0.015 |
| OCM - Hypovolemia/volume depletion ; n (%)* OCM - Anemia ; n (%) | 59 (5.5%)<br>190 (17.6%) | 2,625 (5.4%)<br>9,353 (19.3%) | 0.0044<br>-0.0438 | 106 (3.1%)<br>387 (11.4%) | 2,580 (4.0%)<br>9,554 (14.6%) | -0.0487<br>-0.0953 | 165 (3.7%)<br>577 (12.9%) | 5,205 (4.6%)<br>18,907 (16.6%) | -0.045<br>-0.104 |
| OCM - Dementia ; n (%)* OCM - Depression ; n (%) | 73 (6.8%)<br>204 (18.9%) | 3,560 (7.3%)<br>10,201 (21.0%) | -0.0195<br>-0.0526 | 133 (3.9%)<br>301 (8.9%) | 3,059 (4.7%)<br>8,006 (12.3%) | -0.0394<br>-0.1106 | 206 (4.6%)<br>505 (11.3%) | 6,619 (5.8%)<br>18,207 (16.0%) | -0.054<br>-0.137 |
| ORX - Metformin; n (%)* ORX - 1st and 2nd Generation SUs ; n (%) | 129 (12.0%)<br>96 (8.9%) | 5,947 (12.2%)<br>3,353 (6.9%) | -0.0061<br>0.0742 | 312 (9.2%)<br>298 (8.8%) | 6,884 (10.5%)<br>4.753 (7.3%) | -0.0436<br>0.0552 | 441 (9.9%)<br>394 (8.8%) | 12,831 (11.3%)<br>8,106 (7.1%) | -0.045<br>0.063 |
| ORX - Insulins ; n (%) ORX - Other antidiabetic medications use; n (%) | 92 (8.5%)<br>49 (4.5%) | 3,588 (7.4%)<br>2,328 (4.8%) | 0.0407<br>-0.0142 | 198 (5.8%)<br>169 (5.0%) | 4,670 (7.2%)<br>3,897 (6.0%) | -0.0568<br>-0.0439 | 290 (6.5%)<br>218 (4.9%) | 8,258 (7.3%)<br>6,225 (5.5%) | -0.032<br>-0.027 |
| ORX - PPIs or H2RAs use; n (%)* ORX - NSAIDs ; n (%)* | 299 (27.8%)<br>151 (14.0%) | 15,836 (32.6%)<br>7,708 (15.9%) | -0.1047<br>-0.0533 | 1,088 (32.0%)<br>640 (18.8%) | 18,374 (28.2%)<br>10,402 (15.9%) | 0.0829 | 1,387 (31.0%)<br>791 (17.7%) | 34,210 (30.0%)<br>18,110 (15.9%) | 0.022 |
| ORX - Use of opioids ; n (%)* ORX - Use of antipsychotics ; n (%)* ORX - Use of antidepressants ; n (%) | 418 (38.8%)<br>70 (6.5%)<br>409 (38.0%) | 20,336 (41.9%)<br>2,908 (6.0%)<br>19,790 (40.7%) | -0.0632<br>0.0207<br>-0.0553 | 1,337 (39.4%)<br>139 (4.1%)<br>1,183 (34.8%) | 28,226 (43.2%)<br>3,128 (4.8%)<br>24,738 (37.9%) | -0.0772<br>-0.0340<br>-0.0645 | 1,755 (39.2%)<br>209 (4.7%)<br>1.592 (35.6%) | 48,562 (42.7%)<br>6,036 (5.3%)<br>44,528 (39.1%) | -0.071<br>-0.028<br>-0.072 |
| ORX - Use of anticonyulants : n (%) ORX - Use of anticonyulants : n (%)* | 116 (10.8%)<br>207 (19.2%) | 5,649 (11.6%)<br>10,715 (22.1%) | -0.0254<br>-0.0717 | 388 (11.4%)<br>474 (14.0%) | 8,447 (12.9%)<br>10,973 (16.8%) | -0.0459<br>-0.0776 | 504 (11.3%)<br>681 (15.2%) | 14,096 (12.4%)<br>21.688 (19.1%) | -0.034<br>-0.104 |
| ORX - Use of Benzodiazepines ; n (%)* ORX - Use of dementia meds ; n (%)* | 215 (20.0%)<br>37 (3.4%) | 9,605 (19.8%)<br>1,668 (3.4%) | 0.0050 | 875 (25.8%)<br>100 (2.9%) | 16,742 (25.7%)<br>2,021 (3.1%) | 0.0023<br>-0.0117 | 1,090 (24.4%)<br>137 (3.1%) | 26,347 (23.1%)<br>3,689 (3.2%) | 0.031<br>-0.006 |
| ORX - Use of antiparkinsonian meds ; n (%)* ORX - Use of oral anticoagulants ; n (%)* | 47 (4.4%)<br>122 (11.3%) | 2,335 (4.8%)<br>5,383 (11.1%) | -0.0191<br>0.0063 | 108 (3.2%)<br>423 (12.5%) | 2,814 (4.3%)<br>8,094 (12.4%) | -0.0579<br>0.0030 | 155 (3.5%)<br>545 (12.2%) | 5,149 (4.5%)<br>13,477 (11.8%) | -0.051<br>0.012 |
| ORX - Use of antiplatelet agents; n (%)* LFS - Obesity; n (%) | 123 (11.4%)<br>96 (8.9%) | 6,436 (13.2%)<br>5,778 (11.9%) | -0.0548 | 515 (15.2%)<br>130 (3.8%) | 11,431 (17.5%)<br>4,329 (6.6%) | -0.0622 | 638 (14.3%)<br>226 (5.1%) | 17,867 (15.7%) | -0.039 |
| LFS - Alcohol/Drug Abuse or Dependence; n (%) PFT - Spirometry test only; n (%) | 71 (6.6%)<br>213 (19.8%) | 3,750 (7.7%)<br>12,956 (26.7%) | -0.0427<br>-0.1639 | 66 (1.9%)<br>676 (19.9%) | 2,540 (3.9%)<br>20,587 (31.5%) | -0.1194<br>-0.2678 | 137 (3.1%)<br>889 (19.9%) | 6,290 (5.5%)<br>33,543 (29.5%) | -0.119<br>-0.224 |
| PFT - Spirometry test only (Count - 180 days to 31 days before CED) *mean (sd) | 0.24 (0.71) | 0.34 (0.92) | -0.1217 | 0.22 (0.67) | 0.35 (0.87) | -0.1674 | 0.22 (0.68) | 0.35 (0.89) | -0.164 |
| median [IQR] PFT-Spirometry test only (Count - 30 days to CED) * | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | -0.2139 | 0.00 (0.68) | 0.00 (0.89) | 0.000 |
| mean [sd]median [iQR] PFT-Lung volume, Diffuse capacity, pulmonary stress testing (any); n (%) | 0.15 (0.63)<br>0.00 [0.00, 0.00]<br>151 (14.0%) | 0.21 (0.70)<br>0.00 [0.00, 0.00]<br>9,997 (20.6%) | -0.0901<br>0.0000<br>-0.1752 | 0.11 (0.44)<br>0.00 [0.00, 0.00]<br>249 (7.3%) | 0.23 (0.66)<br>0.00 [0.00, 0.00]<br>10,616 (16.3%) | -0.2139<br>0.0000<br>-0.2817 | 0.12 (0.49)<br>0.00 (0.49)<br>400 (8.9%) | 0.22 (0.68)<br>0.00 (0.68)<br>20,613 (18.1%) | -0.169<br>0.000<br>-0.272 |
| HCU - Pulmonologist visit (180 to 1 day before CED); n (%) | 30 (2.8%) | 1,080 (2.2%) | 0.0384 | 787 (23.2%) | 20,540 (31.5%) | -0.1870 | 817 (18.3%) | 21,620 (19.0%) | -0.018 |
| HCU - Pulmonologist visit on CED; n (%) HCU - Pulmonologist visit (Number of during CAP) * | 2 (0.2%) | 150 (0.3%) | -0.0200 | 84 (2.5%) | 3,729 (5.7%) | -0.1619 | 086 (1.9%) | 3,879 (3.4%) | -0.093 |
| mean (sd)median (lQR) HCU- Number of Internal Medicine/Family Medicine Visits | 0.25 (2.12)<br>0.00 [0.00, 0.00] | 0.17 (1.85)<br>0.00 [0.00, 0.00] | 0.0402 | 0.90 (2.40)<br>0.00 [0.00, 0.00] | 1.43 (3.17)<br>0.00 [0.00, 1.00] | -0.1885<br>0.0000 | 0.74 (2.34)<br>0.00 (2.34) | 0.89 (2.69)<br>0.00 (2.69) | 0.000 |
| HLU - Number of Internal Medicine/Family Medicine visitsmean (sq)median [QR] | 9.76 (13.79)<br>5.00 (1.00, 12.00) | 12.05 (16.93)<br>7.00 (3.00, 15.00) | -0.1483<br>-0.1295 | 7.86 (13.60)<br>4.00 [0.00, 9.00] | 9.00 (13.56)<br>5.00 (2.00, 11.00) | -0.0839<br>-0.0736 | 8.32 (13.65)<br>4.24 (13.65) | 10.30 (15.09)<br>5.85 (15.09) | -0.138<br>-0.112 |
| HCU - Number of Cardiologist visitsmean (sd) | 2.40 (6.18) | 2.46 (5.82) | -0.0100 | 1.27 (3.79) | 1.74 (4.57) | -0.1120 | 1.54 (4.48) | 2.05 (5.14) | -0.106 |
| median [IQR] HCU - Number of Emergency Department (ED) visits v3 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (4.48) | 0.00 (5.14) | -0.015 |
| mean (sd) | 0.87 (1.95)<br>0.00 [0.00, 1.00] | 0.99 (2.07) | -0.0597<br>0.0000 | 0.69 (3.14) | 0.60 (2.44) | 0.0320 | 0.73 (2.90)<br>0.00 (2.90) | 0.77 (2.29) | -0.015 |

# Appendix B

| HCU - Old hospitalization (-180 days to -31 days before CED); n (%) | 251 (23.3%) | 11,887 (24.5%) | -0.0281 | 1,027 (30.2%) | 20,572 (31.5%) | -0.0281 | 1,278 (28.6%) | 32,459 (28.5%) | 0.002 |
|---|---|---|---|---|---|---|---|---|---|
| HCU - Recent hospitalization (-30 days to CED date) ; n (%) | 28 (2.6%) | 2,193 (4.5%) | -0.1028 | 152 (4.5%) | 3,447 (5.3%) | -0.0371 | 180 (4.0%) | 5,640 (5.0%) | -0.048 |
| HCU - Number of hospitalizations during CAP | | | | | | | | | |
| mean (sd) | 0.35 (0.79) | 0.38 (0.78) | -0.0382 | 0.42 (0.73) | 0.44 (0.73) | -0.0274 | 0.40 (0.74) | 0.41 (0.75) | -0.013 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (0.74) | 0.00 (0.75) | 0.000 |
| HCU - Blood eosinophilia or Serum IgE test order; n (%)* | 10 (0.9%) | 418 (0.9%) | 0.0000 | 21 (0.6%) | 461 (0.7%) | -0.0124 | 031 (0.7%) | 879 (0.8%) | -0.012 |
| HCU - Pneumococcal vaccine; n (%) | 133 (12.3%) | 7,651 (15.7%) | -0.0981 | 118 (3.5%) | 4,286 (6.6%) | -0.1419 | 251 (5.6%) | 11,937 (10.5%) | -0.181 |
| HCU - Flu vaccine ; n (%) | 192 (17.8%) | 10,097 (20.8%) | -0.0761 | 368 (10.8%) | 8,600 (13.2%) | -0.0739 | 560 (12.5%) | 18,697 (16.4%) | -0.111 |
| HCU - Bone mineral density ; n (%) | 31 (2.9%) | 2,136 (4.4%) | -0.0801 | 59 (1.7%) | 1,728 (2.6%) | -0.0621 | 090 (2.0%) | 3,864 (3.4%) | -0.086 |
| HCU - Pap smear ; n (%) | 40 (3.7%) | 1,243 (2.6%) | 0.0630 | 113 (3.3%) | 2,079 (3.2%) | 0.0056 | 153 (3.4%) | 3,322 (2.9%) | 0.029 |
| HCU - Mammogram ; n (%) | 120 (11.1%) | 4,993 (10.3%) | 0.0259 | 350 (10.3%) | 5,340 (8.2%) | 0.0725 | 470 (10.5%) | 10,333 (9.1%) | 0.047 |
| HCU - Prostate exam for DRE ; n (%) | 35 (3.2%) | 1,790 (3.7%) | -0.0274 | 28 (0.8%) | 1,170 (1.8%) | -0.0884 | 063 (1.4%) | 2,960 (2.6%) | -0.086 |
| HCU - Number of Echocardiogram * | | | | | | | | | |
| mean (sd) | 0.64 (3.49) | 0.61 (2.97) | 0.0093 | 0.43 (1.23) | 0.47 (1.13) | -0.0339 | 0.48 (2.02) | 0.53 (2.12) | -0.024 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (2.02) | 0.00 (2.12) | 0.000 |
| HCU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy ; n (%) | 60 (5.6%) | 2,516 (5.2%) | 0.0177 | 201 (5.9%) | 4,071 (6.2%) | -0.0126 | 261 (5.8%) | 6,587 (5.8%) | 0.000 |
| HCU - Number of Distinct Medication Prescriptions (not generalized to generics) | | | | | | | | | |
| mean (sd) | 29.01 (22.72) | 28.46 (20.95) | 0.0252 | 26.91 (17.53) | 25.81 (17.21) | 0.0633 | 27.42 (18.91) | 26.94 (18.90) | 0.025 |
| median [IQR] | 23.00 [14.00, 37.00] | 24.00 [14.00, 37.00] | -0.0458 | 23.00 [15.00, 34.50] | 22.00 [14.00, 34.00] | 0.0576 | 23.00 (18.91) | 22.85 (18.90) | 0.008 |
| SES - Copay for pharmacy cost (charges in U.S. \$) | | | | | | | | | |
| mean (sd) | 33.09 (30.71) | 29.56 (35.50) | 0.1064 | 26.74 (27.26) | 24.27 (23.93) | 0.0963 | 28.27 (28.13) | 26.53 (29.43) | 0.060 |
| median [IQR] | 27.02 [12.96, 42.81] | 21.96 [7.85, 38.52] | 0.1524 | 21.25 [9.33, 35.86] | 19.90 [9.93, 32.60] | 0.0526 | 22.64 (28.13) | 20.78 (29.43) | 0.065 |
| SES - Business type | | | | | | | | | |
| Commercial; n (%) | 394 (36.6%) | 11,001 (22.6%) | 0.3104 | | | | 394 (36.6%) | 11,001 (22.6%) | 0.310 |
| Medicare; n (%) | 683 (63.4%) | 37,580 (77.4%) | -0.3104 | | | | 683 (63.4%) | 37,580 (77.4%) | -0.310 |
| SES - Low income indicator ; n (%) | 184 (17.1%) | 12,414 (25.6%) | -0.2086 | | | | 184 (17.1%) | 12,414 (25.6%) | -0.209 |
| SES - Insurance Plan type | | | | | | | | | |
| Comprehensive; n (%) | | | | 1,232 (36.3%) | 21,355 (32.7%) | 0.0758 | 1,232 (36.3%) | 21,355 (32.7%) | 0.076 |
| HMO; n (%) | | | | 959 (28.2%) | 7,748 (11.9%) | 0.4158 | 959 (28.2%) | 7,748 (11.9%) | 0.416 |
| PPO; n (%) | | | | 961 (28.3%) | 28,886 (44.3%) | -0.3374 | 961 (28.3%) | 28,886 (44.3%) | -0.337 |
| Others; n (%) | | | | 245 (7.2%) | 7,275 (11.1%) | -0.1356 | 245 (7.2%) | 7,275 (11.1%) | -0.136 |

<sup>\*</sup> Not included in PS model

**MATCHED** 

| MATCHED | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Number of patients | Referent - Salmeterol<br>1.073 | OPTUM<br>Exposure - Tiotropium<br>1.073 | | Referent - Salmeterol<br>3.285 | MARKETSCAN Exposure - Tiotropium 3 285 | | Referent - Salmeterol | POOLED Exposure - Tiotropium 4 358 | |
| Number of patients Calendar Time - Year of Initiation (2004 - 2020)2004-2006; n (%) | 298 (27.8%) | 303 (28.2%) | -0.0089 | 1,849 (56.3%) | 1,872 (57.0%) | -0.0141 | 2,147 (49.3%) | 2,175 (49.9%) | -0.012 |
| 2007-2008; n (%)<br>2009-2011; n (%) | 103 (9.6%)<br>171 (15.9%) | 87 (8.1%)<br>185 (17.2%) | 0.0528<br>-0.0350 | 403 (12.3%)<br>543 (16.5%) | 376 (11.4%)<br>537 (16.3%) | 0.0278<br>0.0054 | 506 (11.6%)<br>714 (16.4%) | 463 (10.6%)<br>722 (16.6%) | 0.032<br>-0.005 |
| 2012-2015; n (%)<br>2016-2018; n (%)<br>2019-Msr. 2020; n (%) | 157 (14.6%)<br>250 (23.3%)<br>94 (8.8%) | 152 (14.2%)<br>254 (23.7%)<br>92 (8.6%) | 0.0114<br>-0.0094<br>0.0071 | 315 (9.6%)<br>175 (5.3%) | 348 (10.6%)<br>152 (4.6%) | -0.0332<br>0.0323 | 472 (10.8%)<br>425 (9.8%)<br>94 (8.8%) | 500 (11.5%)<br>406 (9.3%)<br>92 (8.6%) | -0.022<br>0.017<br>0.007 |
| DMG - Age | 34(0.000) | 32 (0.0%) | | | | | | | |
| mean (sd)median [IQR] | 69.32 (10.77)<br>70.00 [62.00, 77.00] | 69.31 (10.55)<br>70.00 [62.00, 78.00] | 0.0009 | 70.76 (10.81)<br>72.00 [63.00, 79.00] | 70.58 (10.61)<br>71.00 [63.00, 79.00] | 0.0168<br>0.0934 | 70.41 (10.80)<br>71.51 (10.80) | 70.27 (10.60)<br>70.75 (10.60) | 0.013<br>0.071 |
| DMG - Gender<br>Male; n (%)<br>Female; n (%) | 509 (47.4%)<br>564 (52.6%) | 496 (46.2%)<br>577 (53.8%) | 0.0241 | 1,517 (46.2%)<br>1,768 (53.8%) | 1,528 (46.5%)<br>1,757 (53.5%) | -0.0060<br>0.0060 | 2,026 (46.5%)<br>2,332 (53.5%) | 2,024 (46.4%)<br>2,334 (53.6%) | 0.002 |
| DMG - Gegraphic regionNortheast; n (%) | 100 (9.3%) | 99 (9.2%) | 0.0035 | 348 (10.6%) | 331 (10.1%) | 0.0164 | 448 (10.3%) | 430 (9.9%) | 0.013 |
| South; n (%)North Central; n (%) | 384 (35.8%)<br>276 (25.7%) | 379 (35.3%)<br>265 (24.7%) | 0.0104<br>0.0230<br>-0.0349 | 845 (25.7%)<br>1,107 (33.7%) | 859 (26.1%)<br>1,095 (33.3%) | -0.0091<br>0.0085<br>-0.0087 | 1,229 (28.2%)<br>1,383 (31.7%) | 1,238 (28.4%)<br>1,360 (31.2%)<br>1,330 (30.5%) | 0.011 |
| West; n (%) DRS Combined comorbidity score, 180 daysmean (sd) | 313 (29.2%)<br>2.37 (2.54) | 330 (30.8%)<br>2.30 (2.47) | 0.0349 | 985 (30.0%) | 1,000 (30.4%) | 0.0087 | 1,298 (29.8%) | 1,330 (30.5%) | -0.015 |
| median [IQR] DRS - Frailty Score: Empirical Version (mean) | 2.00 [1.00, 3.00] | 1.00 [1.00, 3.00] | 0.3992 | 1.00 [1.00, 3.00] | 1.00 [1.00, 2.00] | 0.0000 | 1.25 (2.06) | 1.00 (2.01) | 0.123 |
| mean (sd)median [iCR] | 0.21 (0.07)<br>0.19 [0.16, 0.24] | 0.21 (0.07)<br>0.19 [0.16, 0.24] | 0.0000 | 0.19 (0.06)<br>0.18 [0.14, 0.22] | 0.19 (0.06)<br>0.18 [0.14, 0.22] | 0.0000 | 0.19 (0.06)<br>0.18 (0.06) | 0.19 (0.06)<br>0.18 (0.06) | 0.000 |
| PLM - Smoking ; n (%) PLM - Pneumonia ; n (%) | 302 (28.1%)<br>120 (11.2%) | 287 (26.7%)<br>123 (11.5%) | 0.0314 | 319 (9.7%)<br>350 (10.7%) | 329 (10.0%)<br>372 (11.3%) | -0.0101<br>-0.0192 | 621 (14.2%)<br>470 (10.8%) | 616 (14.1%)<br>495 (11.4%) | 0.003<br>-0.019 |
| PLM - Alpha-1 antitrypsin def/Pneumoconioses & other lung disease/Pul fibrosis; n (%) PLM - Oxygen usage; n (%) | 78 (7.3%)<br>155 (14.4%) | 93 (8.7%)<br>161 (15.0%) | -0.0516<br>-0.0169 | 152 (4.6%)<br>575 (17.5%) | 144 (4.4%)<br>623 (19.0%) | 0.0096<br>-0.0388 | 230 (5.3%)<br>730 (16.8%) | 237 (5.4%)<br>784 (18.0%) | -0.004<br>-0.032 |
| PLM - Respiratory arrest/dependence on oxygen; n (%) PLM - CIPAP/BIPAP use; n (%) | 129 (12.0%)<br>63 (5.9%) | 123 (11.5%)<br>57 (5.3%) | 0.0155<br>0.0261<br>0.0748 | 223 (6.8%)<br>129 (3.9%) | 228 (6.9%)<br>144 (4.4%) | -0.0040<br>-0.0251<br>-0.0366 | 352 (8.1%)<br>192 (4.4%)<br>015 (0.3%) | 351 (8.1%)<br>201 (4.6%)<br>015 (0.3%) | -0.010<br>-0.000 |
| PLM - Pulmonary rehabilitation ; n (%)* PLM - Moderate COPD exacerbation - [Count with 365 to 181 days before CED]*mean (x) | 7 (0.7%) | 2 (0.2%) | -0.0648 | 8 (0.2%)<br>1.55 (3.69) | 13 (0.4%) | 0.0195 | 1.58 (3.86) | 1.64 (5.41) | -0.013 |
| median [ICR] PLM - Moderate COPD exacerbation - [Count 180 to 31 days before CED]* | 0.00 [0.00, 1.11] | 0.06 [0.00, 1.57] | -0.0085 | 0.10 [0.00, 1.28] | 0.05 [0.00, 1.22] | 0.0139 | 0.08 (3.86) | 0.05 (5.41) | 0.006 |
| median [IGR] PLM-Moderate COPD exacerbation - [Count with 30 days to CED]* | 1.73 (3.97)<br>0.64 [0.01, 1.83] | 1.77 (6.49)<br>0.62 [0.02, 1.60] | -0.0074<br>0.0037 | 1.29 (2.41)<br>0.54 [0.00, 1.36] | 1.31 (2.33)<br>0.54 [0.00, 1.52] | 0.0084 | 1.40 (2.87)<br>0.56 (2.87) | 1.42 (3.80)<br>0.56 (3.80) | -0.006<br>0.000 |
| mean (sd)median (IQR) | 0.29 (1.12)<br>0.00 [0.00, 0.00] | 0.29 (1.32)<br>0.00 [0.00, 0.00] | 0.0000 | 0.16 (0.54)<br>0.00 [0.00, 0.00] | 0.18 (0.55)<br>0.00 [0.00, 0.00] | -0.0367<br>0.0000 | 0.19 (0.73)<br>0.00 (0.73) | 0.21 (0.81)<br>0.00 (0.81) | -0.026<br>0.000 |
| PLM - Moderate exacerbations ≈1 in 365 days before CED; n (%) PLM - Moderate exacerbations ≈2 in 365 days before CED; n (%) | 861 (80.2%)<br>574 (53.5%) | 872 (81.3%)<br>565 (52.7%) | -0.0279<br>0.0160 | 2,449 (74.6%)<br>1,570 (47.8%) | 2,496 (76.0%)<br>1,617 (49.2%) | -0.0325<br>-0.0280 | 3,310 (76.0%)<br>2,144 (49.2%) | 3,368 (77.3%)<br>2,182 (50.1%) | -0.031<br>-0.018 |
| PLM: Severe COPD exacerbation - [Count with 365 to 181 days before CED] *mean (sd)median [OR] | 0.04 (0.20) | 0.05 (0.25) | -0.0442<br>0.0000 | 0.06 (0.25) | 0.07 (0.27) | -0.0384 | 0.06 (0.24)<br>0.00 (0.24) | 0.07 (0.27)<br>0.00 (0.27) | -0.039 |
| median [QR] PLM - Severe COPD exacerbation - [Count with 180 to 31 days before CED] *mean [sd] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0894 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.06 (0.23) | 0.06 (0.22) | 0.000 |
| median [ICR] PLM - Severe COPD exacerbation - [Count with 30 days lookback] * | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.23) | 0.00 (0.22) | 0.000 |
| mean [dd]median [iQR] PLM - Severe exacerbations >=1 in 365 days before CED; n (%) | 0.01 (0.09)<br>0.00 [0.00, 0.00]<br>106 (9.9%) | 0.01 (0.09)<br>0.00 [0.00, 0.00]<br>106 (9.9%) | 0.0000 | 0.01 (0.06)<br>0.00 (0.00, 0.00)<br>419 (12.8%) | 0.01 (0.09)<br>0.00 [0.00, 0.00]<br>431 (13.1%) | 0.0000<br>0.0000<br>-0.0089 | 0.01 (0.07)<br>0.00 (0.07)<br>525 (12.0%) | 0.01 (0.09)<br>0.00 (0.09)<br>537 (12.3%) | 0.000<br>0.000<br>-0.009 |
| PLM - Sever exect bations -1 in 365 days before CED; n (%) PLM -Governor (%) PLM -Governor (%) | 15 (1.4%)<br>435 (40.5%) | 14 (1.3%)<br>424 (39.5%) | 0.0087 | 63 (1.9%)<br>1,569 (47.8%) | 75 (2.3%)<br>1,636 (49.8%) | -0.0279<br>-0.0400 | 078 (1.8%)<br>2,004 (46.0%) | 089 (2.0%)<br>2,060 (47.3%) | -0.005<br>-0.015<br>-0.026 |
| PRX - LABA (except salmeterol) inhalers; n (%) | 62 (5.8%) | 61 (5.7%) | 0.0043 | 194 (5.9%) | 221 (6.7%) | -0.0329<br>0.0601 | 256 (5.9%)<br>028 (0.6%) | 282 (6.5%)<br>011 (0.3%) | -0.025<br>0.045 |
| PRX - LAMA (except totropium) inhalers; n (%) * PRX - ICS only inhalers; n (%) PRX - LABA/LAMA inhaler use; n (%) * | 14 (1.3%)<br>415 (38.7%)<br>17 (1.6%) | 9 (0.8%)<br>401 (37.4%)<br>8 (0.7%) | 0.0268 | 14 (0.4%)<br>1,534 (46.7%)<br>2 (0.1%) | 2 (0.1%)<br>1,558 (47.4%)<br>3 (0.1%) | -0.0140<br>0.0000 | 1,949 (44.7%)<br>019 (0.4%) | 1,959 (45.0%)<br>011 (0.3%) | -0.006<br>0.017 |
| PRX - LBAP/ICS inhaler use; n (%) PRX - COPD Maintenance therapy inhalers; n (%) | 45 (4.2%)<br>126 (11.7%) | 51 (4.8%)<br>127 (11.8%) | -0.0289 | 107 (3.3%)<br>235 (7.2%) | 110 (3.3%)<br>265 (8.1%) | 0.0000 | 152 (3.5%)<br>361 (8.3%) | 161 (3.7%)<br>392 (9.0%) | -0.011<br>-0.025 |
| PRX - SAMA inhaler use; n (%) PRX - SABA use; n (%) | 108 (10.1%)<br>521 (48.6%) | 115 (10.7%)<br>510 (47.5%) | -0.0197<br>0.0220 | 565 (17.2%)<br>1,486 (45.2%) | 610 (18.6%)<br>1,530 (46.6%) | -0.0365<br>-0.0281 | 673 (15.4%)<br>2,007 (46.1%) | 725 (16.6%)<br>2,040 (46.8%) | -0.033<br>-0.014 |
| PRX - SABA/SAMA use; n (%) PRX - Antibiotics treatment (180 days to 31 days before CED); n (%) PRX - Antibiotics treatment (30 days to CED); n (%) | 242 (22.6%)<br>509 (47.4%)<br>150 (14.0%) | 241 (22.5%)<br>517 (48.2%)<br>157 (14.6%) | 0.0024<br>-0.0160<br>-0.0171 | 817 (24.9%)<br>1,646 (50.1%)<br>450 (13.7%) | 880 (26.8%)<br>1,659 (50.5%)<br>454 (13.8%) | -0.0434<br>-0.0080<br>-0.0029 | 1,059 (24.3%)<br>2,155 (49.4%)<br>600 (13.8%) | 1,121 (25.7%)<br>2,176 (49.9%)<br>611 (14.0%) | -0.032<br>-0.010<br>-0.006 |
| PRX - Systemic Corticosteroids (with CPT) use (180 to 31 days before CED); n (%) PRX - Systemic Corticosteroids (with CPT) use (30 days to CED); n (%) | 537 (50.0%)<br>100 (9.3%) | 540 (50.3%)<br>91 (8.5%) | -0.0060<br>0.0281 | 1,582 (48.2%)<br>365 (11.1%) | 1,592 (48.5%)<br>352 (10.7%) | -0.0060<br>0.0128 | 2,119 (48.6%)<br>465 (10.7%) | 2,132 (48.9%)<br>443 (10.2%) | -0.006<br>0.016 |
| PRX - Roflumilast; n (%) * | 7 (0.7%) | 1 (0.1%) | 0.0952 | 5 (0.2%) | 6 (0.2%) | 0.0000 | 012 (0.3%) | 007 (0.2%) | 0.020 |
| CVD - Unstable angina/M; n (%) CVD - Stable Angina ; n (%) CVD - Any Heart fallure (HF) ; n (%) | 86 (8.0%)<br>46 (4.3%)<br>182 (17.0%) | 78 (7.3%)<br>45 (4.2%)<br>180 (16.8%) | 0.0263<br>0.0050<br>0.0053 | 216 (6.6%)<br>92 (2.8%)<br>501 (15.3%) | 205 (6.2%)<br>71 (2.2%)<br>489 (14.9%) | 0.0163<br>0.0384<br>0.0112 | 302 (6.9%)<br>138 (3.2%)<br>683 (15.7%) | 283 (6.5%)<br>116 (2.7%)<br>669 (15.4%) | 0.016<br>0.030<br>0.008 |
| CVD - Atrial Berillation; n (%) CVD - Other dysrythmias; n (%)* | 143 (13.3%)<br>189 (17.6%) | 140 (13.0%)<br>155 (14.4%) | 0.0089 | 381 (11.6%)<br>344 (10.5%) | 361 (11.0%)<br>368 (11.2%) | 0.0190 | 524 (12.0%)<br>533 (12.2%) | 501 (11.5%)<br>523 (12.0%) | 0.016 |
| CVD - Valve disorder ; n (%) CVD - Implantable cardioverter defibrillator ; n (%)* | 34 (3.2%)<br>14 (1.3%) | 30 (2.8%)<br>22 (2.1%) | 0.0235<br>-0.0619 | 71 (2.2%)<br>32 (1.0%) | 76 (2.3%)<br>36 (1.1%) | -0.0067<br>-0.0098 | 105 (2.4%)<br>046 (1.1%) | 106 (2.4%)<br>058 (1.3%) | 0.000<br>-0.018 |
| CVD - CABG/PCI; n (%) CVD - Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) CVD - Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 74 (6.9%)<br>268 (25.0%)<br>60 (5.6%) | 59 (5.5%)<br>247 (23.0%)<br>66 (6.2%) | 0.0581<br>0.0468<br>-0.0255 | 136 (4.1%)<br>693 (21.1%)<br>163 (5.0%) | 127 (3.9%)<br>657 (20.0%)<br>159 (4.8%) | 0.0102<br>0.0272<br>0.0093 | 210 (4.8%)<br>961 (22.1%)<br>223 (5.1%) | 186 (4.3%)<br>904 (20.7%)<br>225 (5.2%) | 0.024<br>0.034<br>-0.005 |
| CVD - Stroke/TIA ; n (%) CVD - Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) CVD - Hyperlipidemia ; n (%) | 112 (10.4%)<br>514 (47.9%) | 105 (9.8%)<br>511 (47.6%) | 0.0199 | 209 (6.4%)<br>690 (21.0%) | 218 (6.6%)<br>681 (20.7%) | -0.0081<br>0.0074 | 321 (7.4%)<br>1,204 (27.6%) | 323 (7.4%)<br>1,192 (27.4%) | 0.000 |
| CVD - Hypertension; n (%) | 692 (64.5%) | 704 (65.6%) | -0.0231 | 1,347 (41.0%) | 1,335 (40.6%) | 0.0081 | 2,039 (46.8%) | 2,039 (46.8%) | 0.000 |
| CRX - ACE or ARB; n (%) CRX - Mineralocorticold receptor antagonist; n (%) CRX - Loso or Thiaside diuretics: n (%) | 456 (42.5%)<br>43 (4.0%)<br>373 (34.8%) | 471 (43.9%)<br>39 (3.6%)<br>389 (36.3%) | -0.0283<br>0.0209<br>-0.0313 | 1,404 (42.7%)<br>156 (4.7%)<br>1,326 (40.4%) | 1,370 (41.7%)<br>153 (4.7%)<br>1.310 (39.9%) | 0.0202<br>0.0000<br>0.0102 | 1,860 (42.7%)<br>199 (4.6%)<br>1,699 (39.0%) | 1,841 (42.2%)<br>192 (4.4%)<br>1,699 (39.0%) | 0.010<br>0.010<br>0.000 |
| CRX - Statins and other lipid lowering agents; n (%) CRX - Beta blockers; n (%) | 486 (45.3%)<br>341 (31.8%) | 473 (44.1%)<br>324 (30.2%) | 0.0241 | 1,462 (44.5%)<br>937 (28.5%) | 1,412 (43.0%)<br>909 (27.7%) | 0.0302<br>0.0178 | 1,948 (44.7%)<br>1,278 (29.3%) | 1,885 (43.3%)<br>1,233 (28.3%) | 0.028 |
| CRX - CCB and other antihypertensives; n (%) CRX - Digoxin ; n (%)* | 334 (31.1%)<br>52 (4.8%) | 338 (31.5%)<br>51 (4.8%) | -0.0086<br>0.0000 | 1,107 (33.7%)<br>297 (9.0%) | 1,123 (34.2%)<br>283 (8.6%) | -0.0106<br>0.0141 | 1,441 (33.1%)<br>349 (8.0%) | 1,461 (33.5%)<br>334 (7.7%) | -0.008<br>0.011 |
| CRX - Nitrates; n (%)* OCM - Type 1 or 2 DM; n (%) | 100 (9.3%)<br>288 (26.8%) | 90 (8.4%) | 0.0317 | 421 (12.8%)<br>660 (20.1%) | 386 (11.8%)<br>665 (20.2%) | -0.0025 | 521 (12.0%)<br>948 (21.8%) | 476 (10.9%)<br>942 (21.6%) | 0.035 |
| OCM - Occurrence of Diabetic retinopathy/nephropathy/neuropathy; n (%)* OCM - Hypertensive nephropathy; n (%)* | 91 (8.5%)<br>81 (7.5%) | 104 (9.7%)<br>79 (7.4%) | -0.0417<br>0.0038 | 123 (3.7%)<br>100 (3.0%) | 115 (3.5%)<br>86 (2.6%) | 0.0107<br>0.0242 | 214 (4.9%)<br>181 (4.2%) | 219 (5.0%)<br>165 (3.8%) | -0.005<br>0.020 |
| OCMHypotension; n (%)* OCMHypotension; n (%)* OCMCKD II. III. or V: n (%) | 42 (3.9%)<br>29 (2.7%) | 39 (3.6%)<br>32 (3.0%) | -0.0158<br>-0.0180<br>-0.0175 | 75 (2.3%)<br>56 (1.7%) | 88 (2.7%)<br>27 (0.8%) | -0.0256<br>0.0811<br>-0.0251 | 117 (2.7%)<br>085 (2.0%)<br>173 (4.0%) | 127 (2.9%)<br>059 (1.4%)<br>191 (4.4%) | -0.012<br>0.046<br>-0.020 |
| OCM - HD/PD/ESRD; n (%)* OCM - Otteoporosis; n (%) | 93 (8.7%)<br>16 (1.5%)<br>134 (12.5%) | 99 (9.2%)<br>7 (0.7%)<br>142 (13.2%) | 0.0768 | 80 (2.4%)<br>35 (1.1%)<br>457 (13.9%) | 92 (2.8%)<br>22 (0.7%)<br>458 (13.9%) | 0.0424 | 051 (1.2%)<br>591 (13.6%) | 029 (0.7%) | 0.052 |
| OCM - Sleep apnea ; n (%) OCM - Fractures ; n (%) | 139 (13.0%)<br>68 (6.3%) | 132 (12.3%)<br>67 (6.2%) | 0.0211<br>0.0041 | 232 (7.1%)<br>212 (6.5%) | 258 (7.9%)<br>195 (5.9%) | -0.0304<br>0.0249 | 371 (8.5%)<br>280 (6.4%) | 390 (8.9%)<br>262 (6.0%) | -0.014<br>0.017 |
| OCM - Other Arthritis, Arthropathies and Musculoskeletal Pain ; n (%) OCM - Dorsopathies; n (%) | 461 (43.0%)<br>308 (28.7%) | 449 (41.8%)<br>300 (28.0%) | 0.0243<br>0.0155<br>-0.0516 | 1,056 (32.1%)<br>662 (20.2%) | 1,004 (30.6%)<br>639 (19.5%) | 0.0323<br>0.0176<br>0.0367 | 1,517 (34.8%)<br>970 (22.3%) | 1,453 (33.3%)<br>939 (21.5%) | 0.032<br>0.019<br>0.019 |
| OCM - Gout (acute/chronic) ; n (%)* OCM - Hyperthyroidism ; n (%)* OCM - Hypothyroidism ; n (%)* | 7 (0.7%)<br>3 (0.3%)<br>98 (9.1%) | 13 (1.2%)<br>14 (1.3%)<br>104 (9.7%) | -0.1124<br>-0.0206 | 45 (1.4%)<br>18 (0.5%)<br>208 (6.3%) | 32 (1.0%)<br>17 (0.5%)<br>205 (6.2%) | 0.0000 | 052 (1.2%)<br>021 (0.5%)<br>306 (7.0%) | 045 (1.0%)<br>031 (0.7%)<br>309 (7.1%) | -0.026<br>-0.004 |
| OCM - VTE; n (%)* OCM - GERD; n (%) | 39 (3.6%)<br>202 (18.8%) | 46 (4.3%)<br>186 (17.3%) | -0.0359<br>0.0390 | 111 (3.4%)<br>233 (7.1%) | 99 (3.0%)<br>255 (7.8%) | 0.0227<br>-0.0267 | 150 (3.4%)<br>435 (10.0%) | 145 (3.3%)<br>441 (10.1%) | 0.006 |
| OCM - Cancer; n (%) OCM - Hypovolemia/volume depletion; n (%)* | 150 (14.0%)<br>59 (5.5%)<br>190 (17.7%) | 166 (15.5%)<br>54 (5.0%) | -0.0423<br>0.0224<br>0.0731 | 359 (10.9%)<br>105 (3.2%) | 349 (10.6%)<br>115 (3.5%) | 0.0097<br>-0.0167<br>0.0191 | 509 (11.7%)<br>164 (3.8%)<br>566 (13.0%) | 515 (11.8%)<br>169 (3.9%)<br>517 (11.9%) | -0.003<br>-0.005<br>0.033 |
| OCM - Anemia ; n (%) OCM - Dementia ; n (%) OCM - Depression ; n (%) | 73 (6.8%)<br>204 (19.0%) | 161 (15.0%)<br>93 (8.7%)<br>182 (17.0%) | -0.0711<br>0.0521 | 376 (11.4%)<br>128 (3.9%)<br>291 (8.9%) | 356 (10.8%)<br>148 (4.5%)<br>280 (8.5%) | 0.0191 | 201 (4.6%)<br>495 (11.4%) | 241 (5.5%)<br>462 (10.6%) | -0.041<br>0.026 |
| ORX - Metformin; n (%)* | 129 (12.0%) | 117 (10.9%) | 0.0346 | 300 (9.1%) | 304 (9.3%) | -0.0069 | 429 (9.8%) | 421 (9.7%) | 0.003 |
| ORX - 1st and 2nd Generation SUs ; n (%) ORX - Insulins; n (%) ORX - Other antidiabetic medications use: n (%) | 96 (8.9%)<br>92 (8.6%) | 88 (8.2%)<br>102 (9.5%) | 0.0250<br>-0.0314<br>-0.0583 | 284 (8.6%)<br>190 (5.8%) | 279 (8.5%)<br>199 (6.1%) | 0.0036<br>-0.0127<br>-0.0046 | 380 (8.7%)<br>282 (6.5%)<br>213 (4.9%) | 367 (8.4%)<br>301 (6.9%)<br>232 (5.3%) | 0.011<br>-0.016<br>-0.018 |
| ORX - Other antidiabetic medications use; n (%) ORX - PPIs or H2 RAs use; n (%)* ORX - NSAIDs; n (%)* | 49 (4.6%)<br>299 (27.9%)<br>150 (14.0%) | 63 (5.9%)<br>286 (26.7%)<br>172 (16.0%) | 0.0269<br>-0.0560 | 164 (5.0%)<br>1,054 (32.1%)<br>619 (18.8%) | 169 (5.1%)<br>976 (29.7%)<br>557 (17.0%) | 0.0520 | 1,353 (31.0%)<br>769 (17.6%) | 1,262 (29.0%)<br>729 (16.7%) | 0.044<br>0.024 |
| ORX - Use of opioids ; n (%)* ORX - Use of antipsychotics ; n (%)* | 418 (39.0%)<br>69 (6.4%) | 408 (38.0%)<br>60 (5.6%) | 0.0206 | 1,302 (39.6%)<br>137 (4.2%) | 1,273 (38.8%)<br>143 (4.4%) | 0.0164<br>-0.0099 | 1,720 (39.5%)<br>206 (4.7%) | 1,681 (38.6%)<br>203 (4.7%) | 0.018 |
| ORX - Use of antidepressants ; n (%) ORX - Use of anxiolytic/hypnotics; n (%) ORX - Use of anxiolytic/hypnotics; n (%) | 408 (38.0%)<br>116 (10.8%) | 393 (36.6%)<br>106 (9.9%) | 0.0290 | 1,150 (35.0%)<br>383 (11.7%) | 1,152 (35.1%)<br>380 (11.6%) | 0.0021 | 1,558 (35.8%)<br>499 (11.5%) | 1,545 (35.5%)<br>486 (11.2%) | 0.006 |
| ORX - Use of anticonvoliants ; n (%)* ORX - Use of Benzodiazepines; n (%)* ORX - Use of dementia meds ; n (%)* | 207 (19.3%)<br>214 (19.9%)<br>37 (3.4%) | 215 (20.0%)<br>184 (17.1%)<br>45 (4.2%) | -0.0176<br>0.0722<br>-0.0419 | 462 (14.1%)<br>847 (25.8%)<br>97 (3.0%) | 422 (12.8%)<br>863 (26.3%)<br>125 (3.8%) | 0.0381<br>-0.0114<br>-0.0442 | 669 (15.4%)<br>1,061 (24.3%)<br>134 (3.1%) | 637 (14.6%)<br>1,047 (24.0%)<br>170 (3.9%) | 0.022<br>0.007<br>-0.044 |
| URX - Use of dementia meas ; n (s)* ORX - Use of antiparkin sonian meds ; n (%)* ORX - Use of oral anticoagulants ; n (%)* | 37 (3.4%)<br>46 (4.3%)<br>121 (11.3%) | 45 (4.2%)<br>43 (4.0%)<br>125 (11.6%) | 0.0150<br>-0.0094 | 97 (3.0%)<br>104 (3.2%)<br>416 (12.7%) | 125 (3.8%)<br>115 (3.5%)<br>400 (12.2%) | -0.0167<br>0.0151 | 150 (3.4%)<br>537 (12.3%) | 158 (3.6%)<br>525 (12.0%) | -0.011<br>0.009 |
| ORX - Use of antiplatelet agents ; n (%)* | 123 (11.5%) | 108 (10.1%) | 0.0451 | 506 (15.4%) | 482 (14.7%) | 0.0196 | 629 (14.4%) | 590 (13.5%)<br>236 (5.4%) | -0.026 |
| LFS - Obesity; n (%) LFS - Alcohol/Drug Abuse or Dependence ; n (%) | 95 (8.9%)<br>71 (6.6%) | 115 (10.7%)<br>62 (5.8%) | 0.0332 | 126 (3.8%)<br>64 (1.9%) | 121 (3.7%)<br>59 (1.8%) | 0.0074 | 135 (3.1%) | 121 (2.8%) | 0.018 |
| PFT - Spirometry test only; n (%) PFT - Spirometry test only [Count - 180 days to 31 days before CED] * | 213 (19.9%) | 220 (20.5%) | -0.0149 | 672 (20.5%) | 683 (20.8%) | -0.0074 | 885 (20.3%) | 903 (20.7%) | -0.010 |
| mean (xd)median [IQR] PFT- Spirometry test only (Count - 30 days to CED) * | 0.24 (0.71)<br>0.00 [0.00, 0.00] | 0.28 (0.85) 0.00 [0.00, 0.00] | -0.0511<br>0.0000 | 0.23 (0.68)<br>0.00 [0.00, 0.00] | 0.20 (0.65) | 0.0451<br>0.0000 | 0.23 (0.69)<br>0.00 (0.69) | 0.22 (0.70)<br>0.00 (0.70) | 0.014 |
| PFT - Spirometry test only [Count - 30 days to CED] *mean (sd)median [QR] | 0.15 (0.63)<br>0.00 [0.00, 0.00] | 0.13 (0.53)<br>0.00 [0.00, 0.00] | 0.0344 | 0.11 (0.45)<br>0.00 [0.00, 0.00] | 0.13 (0.47) | -0.0435<br>0.0000 | 0.12 (0.50)<br>0.00 (0.50) | 0.13 (0.49)<br>0.00 (0.49) | -0.020 |
| PFT - Lung volume, Diffuse capacity, pulmonary stress testing (any); n (%) | 149 (13.9%) | 155 (14.4%) | -0.0143 | 242 (7.4%) | 260 (7.9%) | -0.0188 | 391 (9.0%) | 415 (9.5%) | -0.017 |
| HCU - Pulmonologist visit (180 to 1 day before CED); n (%) HCU - Pulmonologist visit no CED); n (%) HCU - Pulmonologist visit (Number of full visit of CAP) * | 30 (2.8%)<br>2 (0.2%) | 26 (2.4%)<br>1 (0.1%) | 0.0251 | 781 (23.8%)<br>84 (2.6%) | 794 (24.2%)<br>87 (2.6%) | 0.0094 | 811 (18.6%)<br>086 (2.0%) | 820 (18.8%)<br>088 (2.0%) | -0.005 |
| HCU - Pulmonologist visit (Number of during CAP) *mean (sd)median (IGR) | 0.26 (2.12)<br>0.00 [0.00, 0.00] | 0.23 (2.09)<br>0.00 [0.00, 0.00] | 0.0143 | 0.92 (2.44) | 0.95 (2.51)<br>0.00 [0.00, 1.00] | -0.0121<br>0.0000 | 0.76 (2.37)<br>0.00 (2.37) | 0.77 (2.41)<br>0.00 (2.41) | -0.004 |
| HCU - Number of Internal Medicine/Family Medicine Visitsmean (sd) | 9.78 (13.81) | 10.82 (17.37) | -0.0663 | 7.74 (13.40) | 7.87 (13.19) | -0.0098 | 8.24 (13.50) | 8.60 (14.33) | -0.026 |
| median (ICR) HCU - Number of Cardiologist visitsmean (sq) | 5.00 [1.00, 12.00] | 6.00 [1.00, 13.00]<br>2.06 (5.10) | -0.0637 | 4.00 [0.00, 9.00] | 4.00 [1.00, 9.00]<br>1.29 (4.06) | 0.0000 | 4.25 (13.50)<br>1.58 (4.52) | 4.49 (14.33)<br>1.48 (4.34) | -0.017 |
| median [ICR] HCU - Number of Emergency Department (ED) visits v3 | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (4.52) | 0.00 (4.34) | 0.000 |
| mean (sd) | 0.87 (1.95) | 0.82 (1.93) | 0.0258 | 0.65 (2.71) | 0.65 (3.32) | 0.0000 | 0.70 (2.54) | 0.69 (3.04) | 0.004 |

# Appendix B

| median (ICR) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (2.54) | 0.00 (3.04) | 0.000 |
|---|---|---|---|---|---|---|---|---|---|
| HCU - Old hospitalization (-180 days to -31 days before CED); n (%) | 251 (23.4%) | 224 (20.9%) | 0.0602 | 999 (30.4%) | 969 (29.5%) | 0.0196 | 1.250 (28.7%) | 1.193 (27.4%) | 0.029 |
| HCU - Recent hospitalization (-30 days to CED date) : n (%) | 28 (2.6%) | 23 (2.1%) | 0.0330 | 147 (4.5%) | 131 (4.0%) | 0.0248 | 175 (4.0%) | 154 (3.5%) | 0.026 |
| HCU - Number of hospitalizations during CAP | | | | 2.1.(1.1.1.) | | | | | |
| mean (sd) | 0.35 (0.79) | 0.32 (0.76) | 0.0387 | 0.42 (0.72) | 0.41(0.72) | 0.0139 | 0.40 (0.74) | 0.39 (0.73) | 0.014 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (0.74) | 0.00 (0.73) | 0.000 |
| HCU - Blood eosinophilia or Serum IgE test order: n (%)* | 10 (0.9%) | 11 (1.0%) | -0.0103 | 20 (0.6%) | 25 (0.8%) | -0.0240 | 030 (0.7%) | 036 (0.8%) | -0.012 |
| HCU - Pneumococcal vaccine; n (%) | 133 (12.4%) | 140 (13.0%) | -0.0180 | 115 (3.5%) | 112 (3.4%) | 0.0055 | 248 (5.7%) | 252 (5.8%) | -0.004 |
| HCU - Flu vaccine ; n (%) | 192 (17.9%) | 178 (16.6%) | 0.0344 | 351 (10.7%) | 334 (10.2%) | 0.0163 | 543 (12.5%) | 512 (11.7%) | 0.025 |
| HCU - Bone mineral density ; n (%) | 31 (2.9%) | 34 (3.2%) | -0.0174 | 58 (1.8%) | 66 (2.0%) | -0.0146 | 089 (2.0%) | 100 (2.3%) | -0.021 |
| HCU - Pap smear ; n (%) | 40 (3.7%) | 49 (4.6%) | -0.0451 | 111 (3.4%) | 124 (3.8%) | -0.0215 | 151 (3.5%) | 173 (4.0%) | -0.026 |
| HCU - Mammogram ; n (%) | 120 (11.2%) | 137 (12.8%) | -0.0493 | 334 (10.2%) | 338 (10.3%) | -0.0033 | 454 (10.4%) | 475 (10.9%) | -0.016 |
| HCU - Prostate exam for DRE; n (%) | 35 (3.3%) | 43 (4.0%) | -0.0373 | 27 (0.8%) | 27 (0.8%) | 0.0000 | 062 (1.4%) | 070 (1.6%) | -0.016 |
| HCU - Number of Echocardiogram * | | | | | | | | | |
| mean (sd) | 0.64 (3.50) | 0.46 (1.79) | 0.0648 | 0.44 (1.24) | 0.44 (1.13) | 0.0000 | 0.49 (2.04) | 0.44 (1.32) | 0.029 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (2.04) | 0.00 (1.32) | 0.000 |
| HCU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy ; n (%) | 60 (5.6%) | 62 (5.8%) | -0.0086 | 194 (5.9%) | 190 (5.8%) | 0.0043 | 254 (5.8%) | 252 (5.8%) | 0.000 |
| HCU - Number of Distinct Medication Prescriptions (not generalized to generics) | | | | | | | | | |
| mean (sd) | 28.97 (22.63) | 29.22 (22.55) | -0.0111 | 26.87 (17.54) | 27.20 (17.32) | -0.0189 | 27.39 (18.92) | 27.70 (18.74) | -0.016 |
| median [IQR] | 23.00 [14.00, 37.00] | 24.00 [14.00, 38.00] | -0.0443 | 23.00 [15.00, 35.00] | 24.00 [15.00, 36.00] | -0.0574 | 23.00 (18.92) | 24.00 (18.74) | -0.053 |
| SES - Copay for pharmacy cost (charges in U.S. \$) | | | | | | | | | |
| mean (sd) | 33.13 (30.75) | 34.27 (37.75) | -0.0331 | 26.28 (26.21) | 26.79 (30.17) | -0.0180 | 27.97 (27.40) | 28.63 (32.20) | -0.022 |
| median [IQR] | 27.07 [12.96, 42.81] | 24.89 [11.22, 44.04] | 0.0633 | 21.02 [9.00, 35.43] | 21.11 [10.00, 36.00] | -0.0032 | 22.51 (27.40) | 22.04 (32.20) | 0.016 |
| SES - Business type | | | | | | | | | |
| Commercial; n (%) | 392 (36.5%) | 404 (37.7%) | -0.0248 | | | | 392 (36.5%) | 404 (37.7%) | -0.025 |
| Medicare; n (%) | 681 (63.5%) | 669 (62.3%) | 0.0248 | | | | 681 (63.5%) | 669 (62.3%) | 0.025 |
| SES - Low income indicator ; n (%) | 183 (17.1%) | 201 (18.7%) | -0.0417 | | | | 183 (17.1%) | 201 (18.7%) | -0.042 |
| SES - Insurance Plan type | | | | | | | | | |
| Comprehensive; n (%) | | | | 1,230 (37.4%) | 1,231 (37.5%) | -0.0021 | 1,230 (37.4%) | 1,231 (37.5%) | -0.002 |
| HMO; n (%) | | | | 854 (26.0%) | 819 (24.9%) | 0.0253 | 854 (26.0%) | 819 (24.9%) | 0.025 |
| PPO; n (%) | | | | 956 (29.1%) | 987 (30.0%) | -0.0197 | 956 (29.1%) | 987 (30.0%) | -0.020 |
| Others; n (%) | 1 | l - | | 245 (7.5%) | 248 (7.5%) | 0.0000 | 245 (7.5%) | 248 (7.5%) | 0.000 |

<sup>\*</sup> Not included in PS model